# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# **ANALYSIS PLAN**

for

# **DMID Protocol 17-0088**

**Study Title:** 

A Phase 1, Three-Part, Randomized, Double-Blind, Single and Multiple Subcutaneous Dose Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of Rezafungin in Healthy Adult Subjects

NCT04117607

Version 1.0

**DATE: 06-JUL-2020** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

### STUDY TITLE

| <b>Protocol Number Code:</b> | DMID Protocol 17-0088 |
|---|---|
| <b>Development Phase:</b> | Phase 1 |
| Products: | Rezafungin and Placebo |
| Form/Route: | Solution/Subcutaneous (SC) or Solution/Intravenous (IV) |
| Indication Studied: | Fungal infections |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| Clinical Trial Initiation Date: | 04DEC2019 |
| Clinical Trial Completion Date: | 11MAY2020 |
| Date of the Analysis Plan: | 06JUL2020 |
| Version Number: | 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE | II |
|---------|------------------------------------------------|-----|
| TABLE O | OF CONTENTS | III |
| LIST OF | ABBREVIATIONS | V |
| 1. | PREFACE | 1 |
| 2. | INTRODUCTION | 2 |
| 2.1. | Purpose of the Analyses | 2 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 3 |
| 3.1. | Study Objectives | 3 |
| 3.2. | Endpoints | 3 |
| 3.3. | Study Definitions and Derived Variables | 3 |
| 3.3.1. | Dose Group | 3 |
| 3.3.2. | Baseline | 3 |
| 3.3.3. | Study Day | 4 |
| 4. | SAMPLE SIZE CONSIDERATIONS | 5 |
| 5. | GENERAL STATISTICAL CONSIDERATIONS | 6 |
| 5.1. | General Principles | 6 |
| 5.2. | Timing of Analyses | 6 |
| 5.3. | Analysis Populations | 6 |
| 5.3.1. | Safety Population | 6 |
| 5.3.2. | PK Analysis Population | 6 |
| 5.3.3. | PK Analysis Subset | 6 |
| 5.4. | Covariates and Subgroups | 7 |
| 5.5. | Missing Data | 7 |
| 5.6. | Interim Analyses and Data Monitoring | |
| 5.7. | Multicenter Studies | 7 |
| 5.8. | Multiple Comparisons/Multiplicity | 7 |
| 6. | STUDY SUBJECTS | 8 |
| 6.1. | Disposition of Subjects | 8 |
| 6.2. | Protocol Deviations | 8 |
| 7. | SAFETY EVALUATION | 9 |
| 7.1. | Demographic and Other Baseline Characteristics | 9 |

### **Table of Contents** (continued) Prior and Concurrent Medical Conditions 9 7.1.1. Prior and Concomitant Medications 9 7.1.2. Measurements of Treatment Compliance 9 7.2. 7.3. Adverse Events 9 7.3.1. 7.3.2. Deaths, Serious Adverse Events and other Significant Adverse Events ......11 7.4. 7.5. 7.6. 7.7. 7.8. 7.9. 8. PHARMACOKINETICS ......15 8.1. 9. 10. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR 11. 12. REFERENCES 21 13. LISTING OF TABLES, FIGURES, AND LISTINGS ......22 APPENDIX 1. TABLE MOCK-UPS......23 APPENDIX 3. LISTINGS MOCK-UPS......91

# LIST OF ABBREVIATIONS

| AE | Advarsa Evant/Advarsa Evnarianaa |
|---|---|
| ALT | Adverse Event/Adverse Experience Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Code |
| AUC | Area under the plasma concentration versus time curve |
| $AUC_{inf}$ | Area under the plasma concentration versus time curve from time 0 to infinite time |
| AUC <sub>last</sub> | Area under the plasma concentration versus time curve from time 0 to the time of the |
| | last quantifiable concentration |
| BA | Bioavailability |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| bpm | Beats per minute |
| BUN | Blood Urea Nitrogen |
| BQL | Below Limit of Quantification |
| CI | Confidence Interval |
| CL | Total clearance |
| CL/F | Apparent clearance |
| C <sub>max</sub> | Maximum measured plasma concentration |
| CSR | Clinical Study Report |
| CV % | Coefficient of Variation |
| DMID | Division of Microbiology and Infectious Diseases |
| ECG | Electrocardiogram |
| GM | Geometric Mean |
| λz | The terminal phase elimination rate constant |
| IV | Intravenous |
| LLOQ | Lower Limit of Quantification |
| MAD | Multiple Ascending Dose |
| Max | Maximum |
| MedDRA® | Medical Dictionary for Regulatory Activities |
| Min | Minimum |
| MOP | Manual of Procedures |
| MTD | Maximum tolerated dose |
| N | Number (typically refers to subjects) |
| NCA | Noncompartmental Analysis |
| PE | Physical Examination |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| PR (interval) | Interval measured from the beginning of the P wave to the beginning of the QRS |
| T IC (IIICI Vai) | complex in the heart's electrical cycle as measured by electrocardiogram |
| PT | Preferred Term |
| PTT | Partial Thromboplastin Time |
| QNS | Quantity Not Sufficient |
| Kin | Quality 110t bulliolett |

# **List of Abbreviations** (continued)

| QRS (interval) | The interval between the Q wave and the S wave in the heart's electrical cycle as |
|---|---|
| | measured by electrocardiogram; principal deflection in the electrocardiogram |
| QT (interval) | A measure of the time between the start of the Q wave and the end of the T wave in |
| | the heart's electrical cycle as measured by electrocardiogram |
| QTc (interval) | A measure of time between the start of the Q wave and the end of the T wave in the |
| | heart's electrical cycle measured by electrocardiogram corrected for heart rate |
| SAD | Single Ascending Dose |
| SAE | Serious Adverse Event/Serious Adverse Experience |
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous |
| SD | Standard Deviation |
| SDTM | Study Day Tabulation Model |
| SOC | System Organ Classes |
| t <sub>1/2</sub> | Terminal phase half-life |
| TFL | Tables, Figures, and Listings |
| $T_{max}$ | Time to reach maximum measured plasma concentration |
| VS | Vital Sign |
| V <sub>z</sub> /F | Volume of distribution |
| WBC | White Blood Cell |
| $\begin{array}{c} SC \\ SD \\ SDTM \\ SOC \\ t_{1/2} \\ TFL \\ T_{max} \\ VS \\ V_z/F \end{array}$ | Subcutaneous Standard Deviation Study Day Tabulation Model System Organ Classes Terminal phase half-life Tables, Figures, and Listings Time to reach maximum measured plasma concentration Vital Sign Volume of distribution |

### 1. PREFACE

The Analysis Plan for "A Phase 1, Three-Part, Randomized, Double-Blind, Single and Multiple Subcutaneous Dose Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of Rezafungin in Healthy Adult Subjects" (DMID Protocol 17-0088) describes and expands upon the statistical information presented in the protocol.

The sponsor terminated the study on 27APR2020 due to safety concerns. No subjects were enrolled into Single Ascending Dose (SAD) Cohort 3 (30 mg) and above, any Multiple Ascending Dose (MAD) cohort, or the Bioavailability (BA) cohort. Accordingly, this SAP describes analyses of data from subjects in SAD Cohort 1 (1 mg) and Cohort 2 (10 mg) only.

Due to early termination of the study, the sponsor confirmed an abbreviated clinical study report (CSR) will be provided. The statistical analysis plan noted in the protocol was not drafted and approved prior to study closure and was therefore deemed by the sponsor as not required. This document includes sufficient description of analyses, definitions, tables, figures, and listings (TFLs) for programming of the abbreviated CSR. Within the TFL mock-ups (Appendices 1, 2, and 3), references to abbreviated CSR sections are included. Any deviation from this SAP in the statistical analysis will be described and justified in the abbreviated CSR.

### 2. INTRODUCTION

# 2.1. Purpose of the Analyses

These analyses will assess the safety of single 1 mg or 10 mg subcutaneous doses of rezafungin given subcutaneously and pharmacokinetics (PK) of a single 10 mg subcutaneous dose.

### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

Refer to Protocol v6.0.

### 3.2. Endpoints

Refer to Protocol v6.0.

### 3.3. Study Definitions and Derived Variables

### 3.3.1. Dose Group

Dose Group defines a grouping of subjects used for statistical analysis, where subjects within a Dose Group received the same dose and dosing schedule under the same fasting status. Note that for data from a subject to be analyzed as part of their Dose Group, the subject must also qualify for inclusion into the respective analysis population (As described in Section 5.3) for that data. Definitions for each Dose Group to be analyzed in the report, and their ordering, are provided in the list below.

- SAD Any Dose: Subjects from SAD cohorts who receive any dose of rezafungin.
- SAD 1 mg: SAD, Cohort 1 subjects receiving 1 mg of active drug.
- SAD 10 mg: SAD, Cohort 2 subjects receiving 10 mg of active drug.
- Placebo: SAD subjects receiving placebo.

The "SAD Any Dose" Dose Group will be included in analyses of safety endpoints only.

#### 3.3.2. Baseline

For clinical laboratory results, and vital sign (VS) measurements, the baseline assessment is the last measurement recorded prior to dosing, except for height, weight, and BMI, which baseline will be defined as the measurements recorded at the initial Screening Visit. For electrocardiogram (ECG) results, baseline is defined as the median of the triplicate measurements taken within 60 minutes of dosing. If multiple triplicate measurements are taken prior to dosing, the median of last set of triplicates will be used as baseline.

Age will be based on age at enrollment. Age at enrollment is an integer value with units of years and is calculated from the subject's enrollment date (ENROLLDT) and birth date (BRTHDT) using the following algorithm.

- If month(ENROLLDT) > month(BRTHDT), then AGE = year(ENROLLDT) year(BRTHDT)
- $\bullet \quad If \ month(ENROLLDT) < month(BRTHDT), \ then \ AGE = year(ENROLLDT) year(BRTHDT) 1 \\$
- If month(ENROLLDT) = month(BRTHDT) and day(ENROLLDT) ≥ day(BRTHDT), then AGE = year(ENROLLDT) year(BRTHDT)
- If month(ENROLLDT) = month(BRTHDT) and day(ENROLLDT) < day(BRTHDT), then AGE = year(ENROLLDT) year(BRTHDT) 1

# **3.3.3. Study Day**

The day that the subject received study product is considered Study Day 1 for each subject. The day prior to dosing is considered Study Day = -1, not Study Day = 0.

### 4. SAMPLE SIZE CONSIDERATIONS

No formal sample-size calculations based on testing a statistical hypothesis were constructed. There will be a total of 86 subjects in this three-part trial, 44 subjects in 6 cohorts will receive rezafungin or placebo via SC injection in Part 1/SAD, 32 subjects in 4 cohorts will receive rezafungin or placebo via SC injection in Part 2/MAD, and 10 subjects will receive rezafungin via both SC and IV injections in Part 3/BA. The number of subjects was selected to allow sufficient evaluation of safety, tolerability, and PK of the various dose regimens, and to be consistent with standards of practice for Phase 1 trials.

### 5. GENERAL STATISTICAL CONSIDERATIONS

# **5.1.** General Principles

Safety and PK data will be summarized by Dose Group, following the order shown in Section 3.3. Summary statistics for continuous data will include the mean, standard deviation (SD), median, minimum value (min), and maximum value (max). Summary statistics for discrete data will include counts and percent and may include confidence intervals (CIs) for the percent. When 95% CIs are given for a percent, Wilson Score CIs will be used. All subjects that are randomized will be included in the summaries of demographics, the Safety Population will be used for summaries of safety endpoints, and PK Population or PK Analysis Subset will be used for summaries of PK endpoints.

Generally, for summaries of safety endpoints, denominators will use the number of subjects in the Safety Population. Denominators for study time points of solicited local reactogenicity symptoms, clinical laboratory results, VS, and ECG results will use the number of subjects with an observed result at the time point for the parameter or symptom. Denominators for the conceptual "Max Severity Post-Baseline" time point for solicited local reactogenicity symptoms, clinical laboratory results, VS, and ECG results will use the number of subjects with an observed result for the parameter obtained post-dose.

The sort order of the listings as is indicated in the Implementation Note for each listing shell (Appendix 3).

# **5.2.** Timing of Analyses

The final analysis will be performed after the clinical and non-clinical databases are locked.

# 5.3. Analysis Populations

A tabular listing (Listing 5) and summary table (Table 3) of all randomized and enrolled subjects excluded from the Safety Population, PK Analysis Population, or PK Analysis Subset will be included in the abbreviated CSR. Although there may be multiple reasons for exclusion from a PK Analysis Population or PK Analysis Subset, only one reason will be counted when summarizing reasons for exclusion from analysis populations. Priority for assigning reasons for exclusions will follow the order listed in Table 3.

### **5.3.1.** Safety Population

All subjects that received any amount of study product will be included in the Safety Population.

### 5.3.2. PK Analysis Population

The PK Analysis Population will consist of all subjects who complete one full (as randomized, according to cohort) rezafungin dose and have one post-dose plasma sample with measurable rezafungin Note that all rezafungin concentration results will be included in listings, including results from placebo subjects.

### 5.3.3. PK Analysis Subset

The PK Analysis Subset will be a subset of the PK Analysis Population and will include all subjects in the PK Analysis Population who completed the PK part of the trial without any protocol violations that would likely affect the PK results and who have evaluable plasma concentration data for rezafungin from which at least a subset of the designated PK parameters can be determined. The statistician will review protocol deviations to determine a list of recommended exclusions due to protocol deviations likely to affect PK. The principal

investigator will review the list prior to unblinding and provide confirmation of any exclusions of subjects due to protocol deviations.

# 5.4. Covariates and Subgroups

The protocol does not define any formal subgroup analyses.

# 5.5. Missing Data

No imputation of missing data is planned.

# 5.6. Interim Analyses and Data Monitoring

No interim analysis was conducted prior to study termination.

### 5.7. Multicenter Studies

This is a single-site study.

# 5.8. Multiple Comparisons/Multiplicity

This is a Phase 1 first-in-human study with multiple primary endpoints. Because analyses of primary endpoints are descriptive rather than hypothesis tests, no adjustments for multiple testing are planned

### 6. STUDY SUBJECTS

# 6.1. Disposition of Subjects

Screened subjects who were ineligible for enrollment in the study (screen failures) or eligible but not enrolled will be summarized by inclusion and exclusion criteria (Table 4). Enrolled subjects who were ineligible for inclusion in analysis populations will be summarized by reason for subject exclusion and Dose Group (Table 3). Individual subject listings of subjects who were excluded from the Safety Population or a PK Analysis Population will be listed (Listing 5).

Subject disposition will be summarized (Table 2), showing the number of subjects who screened, enrolled, received study product, completed all PK blood draws, completed final study visit, and early termination.

Subjects who discontinued dosing or terminated early from the study will be listed (Listing 2).

A flowchart showing the disposition of study subjects will be included (Figure 1). This figure will present the number of subjects screened, enrolled, lost to follow-up, and analyzed, by Dose Group.

### 6.2. Protocol Deviations

A summary of protocol deviations will be presented by deviation category, deviation type, and Dose Group (Table 1). This table will provide both the number of subjects and the number of deviations for each category. All subject-specific protocol deviations and non-subject-specific protocol deviations will be listed (Listing 3 and Listing 4).

### 7. SAFETY EVALUATION

All safety analyses will be performed using the Safety Population.

Any medical condition that is present at the time that the subject is screened will be considered baseline and not reported as an AE unless it worsens in severity or increases in frequency during the study. The denominators for percent values will be indicated within the table or table header and denoted as N. Moreover, events summarized by subject will be coded to the highest severity observed over the indicated time period. Toxicity grading scales for adverse events, solicited reactogenicity symptoms, safety labs, VS, and ECG are provided in the protocol v6.0.

# 7.1. Demographic and Other Baseline Characteristics

Demographic summaries will include all subjects that were randomized. Sex, ethnicity, and race of all subjects will be summarized categorically by Dose Group (Table 5). Age at enrollment and height, weight, and BMI at screening will be summarized as continuous variables by Dose Group (Table 6). Individual subject listings will be presented for all demographic and baseline characteristics (Listing 6).

#### 7.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past pre-existing medical conditions will be MedDRA coded using MedDRA dictionary version 23.0 or higher. Summaries of subjects' pre-existing medical conditions by MedDRA system organ class (SOC) will be presented by Dose Group (Table 7). Individual subject listings will be presented for all medical conditions (Listing 7).

#### 7.1.2. Prior and Concomitant Medications

All medications will be coded using the current version of the WHO Drug dictionary. The use of prior and concomitant medications taken during the study will be summarized by Anatomical Therapeutic Code (ATC) 1 and ATC 2 (separately in Table 33 for prior medications and Table 34 for concomitant medications). Individual subject listings will be presented for all prior and concomitant medications (separately in Listing 23 for prior medications and Listing 24 for concomitant medications).

# **7.2.** Measurements of Treatment Compliance

Date and time of dosing will be presented in Listing 8. Concentration in plasma for Cohort 2 (including placebo) will be presented in Listing 31.

#### 7.3. Adverse Events

When calculating the proportions of subjects with AEs within a given MedDRA category, each subject will only be counted once and any repetitions of AEs within a subject will be ignored, and the event will be reported according to the worst severity recorded (separately for related and unrelated AEs, when both severity and relatedness are tabulated).

### 7.3.1. Solicited Reactogenicity Symptoms

For each solicited local reactogenicity symptom, the number and percentage of subjects reporting each symptom will be summarized by maximum severity for a specified time point and Dose Group.

Maximum severity for each symptom based on functional grading and measurement grading criteria as described in protocol v6.0 will be summarized separately. All pre-dose and post-dose solicited local reactogenicity will be presented in Listing 9.

The following summaries for solicited local reactogenicity symptoms will be presented:

- The number and proportion of subjects with local symptoms, summarized by Dose Group and symptom. A 95% CI will be presented by Dose Group for each local symptom (Table 9).
- The number and proportion of subjects with local symptoms, summarized by Dose Group, symptom, and maximum severity. A 95% CI will be presented by Dose Group for each local symptom (Table 10).
- The number and proportion of subjects with local symptoms, summarized by Dose Group, symptom, time point, and maximum severity (including maximum severity post-baseline) (Table 11).
- By Dose Group, bar charts of proportions of subjects with local symptoms by maximum severity (each subject counted once per symptom) (Figure 2).
- By Dose Group and time point, bar charts of proportions of subjects with each local symptom by maximum severity (starting at Figure 3, continuing through Figure 16).

The following solicited local reactogenicity symptoms will be presented (in order):

• Pain, tenderness, pruritus (itching), ecchymosis (bruising) (functional grade), ecchymosis (bruising) (measurement grade), induration (hardness)/ swelling (functional grade), induration (hardness)/ swelling, (measurement grade), erythema (redness) (functional grade), erythema (redness) (measurement grade), nodule (functional grade), nodule (measurement grade), ulceration (functional grade), and ulceration (measurement grade).

### 7.3.2. Unsolicited Adverse Events

A brief overall summary of AEs by Dose Group including number of subjects with at least one solicited reactogenicity event of any severity, number of subjects with ulceration, number of subjects with at least one AE of any severity, number of subjects with at least one related AE of any severity, and number of subjects with at least one SAE (Table 8).

All AEs will be presented in listings (Listing 10). A subject listing of non-serious AEs of moderate or greater severity will also be reported (Table 15).

The following summaries for unsolicited adverse events will be presented:

- The total number of AEs and the number and proportion of subjects reporting at least one unsolicited AE will be summarized by Dose Group, SOC, and PT. Denominators for percentages are the number of subjects in the Safety Population. A 95% CI will be presented by Dose Group for each SOC and PT (Table 12).
- The number and proportion of subjects reporting at least one AE, summarized by Dose Group, SOC, PT, maximum severity, and relatedness (Table 13).
- By Dose Group, bar charts of proportions of subjects with related serious and non-serious AEs by maximum severity and SOC. This figure describes the number of subjects with an event (each subject counted once per SOC) (Figure 17).

• By Dose Group, bar charts of numbers of related serious and non-serious AEs by severity and SOC. This figure describes the total number of occurrences of each event, including multiple occurrences per subject (Figure 18).

# 7.4. Deaths, Serious Adverse Events and other Significant Adverse Events

Individual data listings of deaths and other SAEs will be provided (Table 14).

# 7.5. Pregnancies

An individual data listing of pregnancy reports will be provided if a pregnancy occurs pose-dosing (Listing 25, Listing 26, Listing 27, Listing 28, Listing 29). Contraceptive method will be listed in Listing 30.

# 7.6. Clinical Laboratory Evaluations

If the time of sample collection for clinical laboratory evaluations was prior to 23DEC2019, then grading will follow toxicity grade criteria from protocol v3.0. If the time of sample collection was on or after 23DEC2019, then grading will follow toxicity grade criteria from protocol v4.0. Note that toxicity ranges from protocol v4.0 through v6.0 were identical.

- CHEM: Total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and triglycerides were removed from clinical lab collection after protocol v3.0.
- COAG: Prothrombin time and activated PTT toxicity ranges were updated after protocol v3.0.
- UA: Blood in urine (microscopic) toxicity ranges were updated after protocol v3.0.

All screening and safety laboratory results will be listed in Listing 11 (CHEM), Listing 12 (HEM), Listing 13 (COAG), Listing 14 (UA), Listing 15 (serology), Listing 16 (urine toxicity), and Listing 17 (pregnancy test). Abnormal laboratory results (laboratory results outside of the normal range on time of collection) will be listed in Table 16 (CHEM), Table 17 (HEM), Table 18 (COAG), and Table 19 (UA).

Laboratory results will be summarized in tables and figures:

- Tabularly, by parameter, Dose Group, time point, and toxicity grade (including maximum severity post-baseline). Summaries will be presented in Table 20 (CHEM), Table 22 (HEM), Table 24 (COAG), and Table 26 (UA). When calculating the proportions of subjects with a laboratory toxicity, each subject will only be counted once per toxicity grade and any repetitions of laboratory toxicities within a subject will be ignored, and the event will be reported according to the worst severity recorded. Parameters with no specified toxicity ranges listed in protocol will be excluded from this summary.
- Tabularly, by summary statistics for change from baseline, reported by parameter, Dose Group, and time point. Summaries will be presented in Table 21 (CHEM), Table 23 (HEM), and Table 25 (COAG).
- Graphically, using box plots of change from baseline by parameter, Dose Group, and time point.
  - o CHEM: Beginning at Figure 19 and continuing through Figure 35.
  - o HEM: Beginning at Figure 36 and continuing through Figure 45.
  - o COAG: Figure 46, Figure 47, and Figure 48.

The following laboratory parameters will be presented (in order):

- Chemistry (CHEM): sodium, potassium, calcium, phosphorus, chloride, total carbon dioxide, glucose, blood urea nitrogen, creatinine, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglycerides, total protein, albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total bilirubin, direct bilirubin, creatine phosphokinase. Total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and triglycerides parameters were removed after Protocol v3.0. Only Cohort 1 subjects have results for the specified parameters. Due to limited number of subjects with available results, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and triglycerides will only be presented in Table 21 and Listing 11 and will be excluded from the change from baseline figures.
- Hematology (HEM): hemoglobin, hematocrit, RBC count, WBC count, neutrophil count, lymphocyte count, monocyte count, eosinophil count, basophil count, platelet count.
- Coagulation (COAG): prothrombin time, activated PTT, INR
- Urinalysis (UA): protein, glucose, occult blood.

By protocol, microscopic evaluation of urine or complete urinalysis is only performed if dipstick urinalysis is positive for blood. If complete UA or microscopic results were obtained in the absence of an abnormal dipstick result (or without dipstick tests being done), results of the complete UA or microscopy will still be summarized. Results determined using both methods will be listed. In tables, dipstick results will be presented prior to complete UA or microscopy results.

Laboratory parameters that have grading criteria for both decreases (result lower than normal range) and increases (result higher than normal range) will be summarized separately by direction of change. For example, sodium will be summarized separately as "Sodium, Decrease" and "Sodium, Increase."

In tables summarizing toxicity grading, maximum severity observed after dosing will be summarized (max severity post-baseline, including unscheduled visits) for each parameter. Results of maximum severity for "Any Parameter" will be included for all clinical laboratory results. For "Any Parameter" results, the maximum severity across all laboratory parameters in the respective category is summarized by time point.

Unscheduled clinical laboratory evaluations will be listed, but excluded from tabular and graphical summaries, except when calculating the maximum severity post-baseline. Any pre-existing abnormal lab results at screening will be graded and presented in listings but will not be reported as an AE unless they are treatment-emergent (i.e. it worsens after dosing, meaning for continuous parameters that an increase toxicity can only be assigned if the result is numerically higher than baseline and a decrease toxicity can only be assigned if the result is numerically lower than baseline.)

# 7.7. Vital Signs and Physical Evaluations

All VS measurements will be presented in Listing 18.

VS will be summarized in tables and figures:

- Tabularly, by parameter, Dose Group, time point, and toxicity grade (including maximum severity post-baseline). Respiratory rate measurements are not graded, and so will not be included in this summary. (Table 27).
- Tabularly, by summary statistics for change from baseline, reported by parameter, Dose Group, and time point. (Table 28).

• Graphically, using box plots of change from baseline by parameter, Dose Group, and time point. (Figure 49, Figure 50, Figure 51, Figure 52, Figure 53).

The following parameters will be reported (in order): systolic blood pressure (BP), diastolic BP, heart rate, respiratory rate, and temperature.

VS parameters that have grading criteria for both decreases (result lower than normal range) and increases (result higher than normal range) will be summarized separately by direction of change. For example, systolic blood pressure will be summarized separately as "Systolic Blood Pressure, Decrease" and "Systolic Blood Pressure, Increase."

In tables summarizing toxicity grading, maximum severity observed after dosing will be summarized for each parameter. Results of maximum severity for "Any Parameter" will also be included. For "Any Parameter" results, the maximum severity across all vital sign parameters is summarized by time point.

Unscheduled VS measurements will be listed, but excluded from tabular and graphical summaries, except when calculating the maximum severity post-baseline. Baseline for height, weight, and BMI will be the measurement taken at Screening Visit, baseline for the rest of the VS parameters is defined as the last vital sign parameter taken before dosing on Day 1 (including any repeats). Repeated VS due to clinic error or technical problem will be used for all analyses instead of the original vital sign result. Additional measurements taken as follow-up for safety will be included in listings and in computing maximum severity post baseline, but not as separate time points in summary tables. For repeats that were done due to delayed dosing, the last measurement prior to dosing will be considered as baseline for that subject.

Abnormal PE findings will be listed in Listing 19.

# 7.8. 12-Lead Standard Electrocardiogram

All 12-lead standard ECG measurement results, overall interpretation, and findings will be listed in Listing 20, Listing 21, and Listing 22.

12-lead standard ECG results will be summarized in tables and figures:

- Tabularly, 12-lead standard ECG change in overall interpretation from baseline will be shown by Dose Group and time point (Table 29).
- Tabularly, by parameter, Dose Group, time point, and toxicity grade (including maximum severity post-baseline) (Table 30).
- Tabularly, by summary statistics for change from baseline, reported by parameter, Dose Group, and time point (Table 31).
- Tabularly, by Dose Group, time point, and sex based on QTcF categories according to the ICH Guideline E14 "Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs" (protocol v6.0 Section 10.5.2). (Table 32).
- Graphically, using box plots of change from baseline by parameter, Dose Group, and time point (Figure 54, Figure 55, Figure 56, Figure 57, Figure 58, Figure 59).

The following parameters will be presented (in order): PR interval, QRS duration, QT interval, QTcF interval, RR interval, and mean ventricular rate.

Unscheduled 12-lead standard ECG measurements will be listed but excluded from tabular and graphical summaries. Individual interval measurements will be presented in listings along with overall interpretation

and comments. Other ECG findings besides interpretation will also be included in listings. Repeated ECG due to clinic error or technical problem will be used for all analyses instead of the original ECG result. Additional ECG measurements taken as follow-up for safety will be included in listings and in computing maximum severity post baseline, but not as separate time points in summary tables. For repeats that were done due to delayed dosing, the median of the last triplicate ECG measurement prior to dosing will be considered as baseline for that subject.

# 7.9. Concomitant Medications

All medications will be coded using the current version of the WHO Drug dictionary. The use of prior and concomitant medications taken during the study will be summarized by ATC 1 and ATC 2 (separately in Table 33 for prior medications and Table 34 for concomitant medications). Individual subject listings will be presented for all prior and concomitant medications (separately in Listing 23 for prior medications and Listing 24 for concomitant medications).

### 8. PHARMACOKINETICS

Time points below the lower limit of quantification (LLOQ), referred to as below limit of quantification (BQL), preceding the first PK concentration above the LLOQ will be imputed as 0 for plotting and for all calculations including NCA and summary statistics. All other BQL values will be missing for analysis purposes. There will be no imputation of missing concentrations. A geometric mean (GM) of concentrations will be treated as missing for sets of data points containing more than 1 BQL value.

Collection of plasma samples outside of the protocol defined time window for the time point will not result in exclusion of the sample result from noncompartmental analysis (NCA). Plasma samples collected out of window will be evaluated on a case-by-case basis. Samples will be considered substantially out of window if PK samples were not collected within  $\pm$  10 min for the 0.5 hour time point,  $\pm$  20 min of the targeted collection time (nominal time point) for time points 12 hours post-dose and earlier and within  $\pm$  1 hour for nominal time points from 24 to 144 hours post-dose, and  $\pm$  2 days on Day 14 and Day 30. Results from substantially out of window samples will be excluded from concentration summary statistics by nominal time points and plots of mean concentration, but included in NCA and in plots of individual concentrations.

Drug concentrations in plasma will be listed for subjects in Cohort 2, including placebo, with BQL and PK analyses-excluded samples indicated and with separate columns for concentrations reported by the lab and concentrations used for analysis (Listing 31). The column containing concentrations reported from the lab may include codes such as "BQL" or "QNS" (Quantity Not Sufficient) while the column containing concentrations used for analysis will contain numeric data only, including imputed values such as zeros for pre-dose timepoints reported as BQL. The listings will also indicate the nominal time (i.e., the planned time) and actual post-dose time in h associated with the sample.

The PK Analysis Subset will be used when summarizing PK concentrations. Summary statistics will be given for rezafungin concentrations by nominal time (Table 35).

Rezafungin concentrations will be also be shown graphically:

- Individual subject concentration-time profiles within 144 hours post-dose (Day 7) with y-axis on the linear scale (Figure 60).
- Individual subject concentration-time profiles within 144 hours post-dose (Day 7) with y-axis on the logarithmic scale (Figure 61).
- Individual subject concentration-time profiles for all time points with y-axis on the linear scale (Figure 62).
- Individual subject concentration-time profiles for all time points with y-axis on the logarithmic scale (Figure 63).
- GM concentration-time profiles within 144 hours post-dose (Day 7) y-axis on the linear scale. Error bars will show the mean  $\pm$  1 SD (Figure 64).
- GM concentration-time profiles within 144 hours post-dose (Day 7) y-axis on the logarithmic scale (Figure 65).
- GM concentration-time profiles for all time points with y-axis on the linear scale. Error bars will show the mean  $\pm$  1 SD (Figure 66).
- GM concentration-time profiles for all time points with y-axis on the logarithmic scale (Figure 67).

### 8.1. Noncompartmental Analysis

PK parameters will be estimated through an NCA using Phoenix<sup>®</sup> WinNonlin<sup>®</sup> version 8.2 or later (Certara, Princeton, NJ). Actual post-dose time will be used for the estimation of PK parameters instead of nominal time. Individual PK parameter estimates will be listed. PK Analysis Subset will be used when summarizing PK parameters. Summary tables including mean, SD, min, max, median, coefficient of variation (CV %), and GM will be presented (Table 36). Definition of CV is provided below.

For an independent identically distributed random sample  $\{x_1, x_2, ..., x_n\}$  from a log-normal distribution, let  $s^2$  be the sample variance statistic of the natural log-transformed values of the sample. The CV was defined as:

$$CV = \sqrt{\exp(s^2) - 1}$$

Phoenix® WinNonlin® NCA will use the following settings to compute parameters from plasma rezafungin concentration data:

- Linear Up Log Down calculation method
- Uniform weighting
- Extravascular Dosing
- Lambda Z Acceptance Criteria
  - Rsq adjusted  $\geq 0.90$
  - Span  $\geq$  3.0 half-lives
  - Includes at least 3 timepoints after T<sub>max</sub>

All estimable PK parameters and terminal phase PK parameters that meet Lambda Z acceptance criteria will be listed in Listing 32. A definition for each PK parameter for the SAD cohorts are defined below.

#### $C_{max}$

Maximum concentration ( $C_{max}$ ) is defined as the maximum observed drug concentration observed over all PK sample concentrations. It will be obtained from the **Cmax** parameter calculated by WinNonlin<sup>®</sup>. If there is no measurable concentration in the subject's PK profile, then  $C_{max}$  will be missing for that subject.  $C_{max}$  will be reported in units of ng/mL.

#### $T_{max}$

Time of maximum concentration  $(T_{max})$  is defined as the time at which the  $C_{max}$  occurs. It will be obtained from the **Tmax** parameter calculated by WinNonlin<sup>®</sup>. If there is no measurable  $C_{max}$  in the subject's PK profile, then  $T_{max}$  will be missing for that subject.  $T_{max}$  will be reported in units of h.

### $\lambda z$

The terminal phase elimination rate constant ( $\lambda z$ ) is defined as the first-order rate constant describing the rate of decrease of drug concentration in the terminal phase (defined as the terminal region of the PK curve where drug concentration follows first-order elimination kinetics).  $\lambda z$  will be computed as the slope of a terminal region consisting of  $\geq 3$  successive points in the plot of log-transformed concentration data versus time.  $\lambda z$  will be estimated using uniform weighting.

Time points used in the estimation of  $\lambda z$  will be initially selected using the WinNonlin<sup>®</sup> automatic algorithm. Manually chosen time points may be used at the discretion of the PK analyst after examination of the automatically chosen points in the context of the semi-log profile. The set of points chosen must contain only

timepoints after  $T_{max}$ , include at least 3 timepoints, and satisfy the Lambda Z Acceptance Criteria described above. Otherwise, the elimination rate constant and all derived parameters (apparent terminal elimination half-life [ $t_{1/2}$ ], AUC Extrapolated to Infinity [AUC<sub>0-inf</sub>], Apparent Clearance [CL/F], Apparent volume of distribution during terminal phase [ $V_z/F$ ]) will be treated as missing.

The range of concentrations used to estimate  $\lambda z$  for each profile will be inspected by the PK analyst, who may adjust the set of concentrations used to estimate  $\lambda z$  if deemed necessary, but manually selected ranges must satisfy the same acceptance criteria as those chosen automatically by the WinNonlin® algorithm. Sets of drug concentrations used to calculate  $\lambda z$  will be indicated in the listing for concentration. This parameter will be obtained from the **Lambda\_z** parameter calculated by WinNonlin®.  $\lambda z$  will be reported in units of 1/h.

#### t<sub>1/2</sub>

The  $t_{1/2}$  is defined as the time required for the drug concentration to decrease by a factor of one-half in the terminal phase. The  $t_{1/2}$  can be estimated as  $\ln(2) / \lambda z$ . It will be obtained from the **HL\_Lambda\_z** parameter calculated by WinNonlin<sup>®</sup>. Half-life will be reported in units of h.

### **AUC**

AUC<sub>0-last</sub> is defined as the area under the concentration-time curve from dosing (time 0) to the time of the last measured concentration. AUC<sub>0-last</sub> will be estimated using the Linear Up Log Down calculation method and obtained from the **AUClast** parameter calculated by WinNonlin<sup>®</sup>.

 $AUC_{0-inf}$  is defined as the total area under the concentration-time curve from dosing (time 0) taken to the limit as the end time becomes arbitrarily large.  $AUC_{0-inf}$  can be calculated by adding  $AUC_{0-last}$  to an extrapolated value equal to the last measured concentration greater than the LLOQ divided by  $\lambda z$ :

$$AUC_{0-\inf} = AUC_{0-last} + \frac{C_{last}}{\lambda z},$$

where  $C_{last}$  is the last measured concentration  $\geq$  LLOQ. AUC<sub>0-inf</sub> will be obtained from the **AUCINF\_obs** parameter calculated by WinNonlin<sup>®</sup>. If the amount extrapolated portion of AUC<sub>0-inf</sub> is >20%, the estimated AUC<sub>0-inf</sub> value will be flagged when listed in the report and will be excluded from statistical summaries of parameter estimates and downstream calculations.

All AUCs will be reported in units of h\*ng/mL.

#### CL/F

Apparent clearance (CL/F) will be computed as Dose/AUC<sub>0-inf</sub>. Clearance will be reported in units of L/h.

#### $V_z/F$

Apparent volume of distribution during terminal phase  $(V_z/F)$  after non-intravenous administration will be calculated as  $(CL/F)/\lambda z$ . Volume will be reported in units of L.

### 9. REPORTING CONVENTIONS

The mean, median, SD, and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Order statistics, such as the min and max, will use the same number of decimal places as the original data. Proportions will be presented as two decimal places; values <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values < 1% will be presented as "<1".

For PK, AUCs will be reported as whole numbers (or using 3 significant digits if less than 100). t1/2, Tmax, CL/F, and Vz/F values will be reported to one decimal place (or to 2 decimal places if less than 1).  $\lambda z$  values will be reported to 3 significant digits. Cmax will be reported to 3 significant digits. The mean, median, SD, and any other statistics other than quantiles will be reported one significant digit greater than the reported data. Order statistics, such as the min and max, will use the same number of significant digits as the original data.

Listings of individual subject data include a Subject ID column. The subject identifiers assigned by site staff are replaced throughout this report with the Study Day Tabulation Model (SDTM) variable USUBJID to protect the confidentiality of those who volunteered to participate in this protocol. USUBJID has been created as a composite of the 3-letter EDC platform code followed by a numeric identifier assigned chronologically to enrolled subjects as well as screening failures across all sites and protocols in the EDC platform. Any data sharing activities will include the USUBJID and not the subject identifiers assigned at the site.

# 10. TECHNICAL DETAILS

SAS version 9.4 or above or R versions 3.2 or above will be used to generate tables, figures, and listings. PK parameters will be estimated through an NCA using Phoenix® WinNonlin® version 8.2 or later (Certara, Princeton, NJ).

# 11. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

The sponsor terminated the study on 27APR2020 due to safety concerns. No subjects were enrolled into SAD Cohort 3 (30 mg) and above, any MAD cohort, or the BA cohort. Only SAD 1 mg and SAD 10 mg Dose Groups will be included in the final safety analysis and SAD 10 mg Dose Group will be included in the final PK analysis.

# 12. REFERENCES

# 13. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3.

# **APPENDICES**

# APPENDIX 1. TABLE MOCK-UPS

# LIST OF TABLES

| Table 1: | Distribution of Protocol Deviations by Category, Type, and Dose Group | 25 |
|---|---|---|
| Table 2: | Subject Disposition by Dose Group | 26 |
| Table 3: | Analysis Populations by Dose Group | 27 |
| Table 4: | Ineligibility Summary of Screen Failures | 28 |
| Table 5: | Summary of Categorical Demographic and Baseline Characteristics by Dose Group | 30 |
| Table 6: | Summary of Continuous Demographic and Baseline Characteristics by Dose Group | 31 |
| Table 7: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Dose Group | 32 |
| Table 8: | Overall Summary of Adverse Events by Dose Group | 33 |
| Table 9: | Number and Percentage of Subjects Experiencing Solicited Reactogenicity Symptoms with 95% Confidence Intervals by Symptom and Dose Group | 34 |
| Table 10: | Number and Percentage of Subjects Experiencing Solicited Reactogenicity Symptoms with 95% Confidence Intervals by Symptom, Severity, and Dose Group | 35 |
| Table 11: | Number and Percentage of Subjects Experiencing Solicited Reactogenicity Symptoms by Symptom, Severity, Time Point, and Dose Group | 37 |
| Table 12: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Dose Group | 38 |
| Table 13: | Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship, and Dose Group | 39 |
| Table 14: | Listing of Serious Adverse Events | 40 |
| Table 15: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | 41 |
| Table 16: | Listing of Abnormal Laboratory Results – Chemistry | 43 |
| Table 17: | Listing of Abnormal Laboratory Results - Hematology | 44 |
| Table 18: | Listing of Abnormal Laboratory Results - Coagulation | 45 |
| Table 19: | Listing of Abnormal Laboratory Results - Urinalysis | 46 |
| Table 20: | Chemistry Toxicity Grade by Parameter, Severity, Dose Group, and Time Point | 47 |

| Table 21: | Chemistry Change from Baseline by Parameter, Dose Group, and Time Point | 48 |
|---|---|---|
| Table 22: | Hematology Toxicity Grade by Parameter, Severity, Dose Group, and Time Point | 49 |
| Table 23: | Hematology Change from Baseline by Parameter, Dose Group, and Time Point | 49 |
| Table 24: | Coagulation Toxicity Grade by Parameter, Dose Group, and Time Point | 50 |
| Table 25: | Coagulation Change from Baseline by Parameter, Dose Group, and Time Point | 50 |
| Table 26: | Urinalysis Toxicity Grade by Parameter, Severity, Dose Group, and Time Point | 51 |
| Table 27: | Vital Sign Toxicity Grade by Parameter, Severity, Dose Group, and Time Point | 52 |
| Table 28: | Vital Sign Change from Baseline by Parameter, Dose Group, and Time Point | 53 |
| Table 29: | ECG Overall Interpretations, Post Dose Compared to Baseline by Dose Group and Time Point | 54 |
| Table 30: | ECG Toxicity Grade by Parameter, Severity, Dose Group, and Time Point | 55 |
| Table 31: | ECG Change from Baseline by Parameter, Dose Group, and Time Point | 56 |
| Table 32: | Summary of QTcF by Dose Group and Time Point | 57 |
| Table 33: | Number and Percentage of Subjects with Prior Medications by WHO Drug<br>Classification and Dose Group | 58 |
| Table 34: | Number and Percentage of Subjects with Concomitant Medications by WHO Drug Classification and Dose Group | 59 |
| Table 35: | Rezafungin Concentrations in Plasma, SAD 10 mg Dose Group | 60 |
| Table 36: | Summary Statistics for Rezafungin PK Parameters in Plasma – SAD 10 mg Dose Group | 61 |

# **10.2** Protocol Deviations

Table 1: Distribution of Protocol Deviations by Category, Type, and Dose Group

| | | Num | Number of Subjects (Number of Deviations) | | |
|---|---|---|---|---|---|
| Category | Deviation Type | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) | All Subjects<br>(N=X) |
| Eligibility/enrollment | Any type | x (x) | x (x) | x (x) | x (x) |
| | Did not meet inclusion criterion | x (x) | x (x) | x (x) | x (x) |
| | Met exclusion criterion | x (x) | x (x) | x (x) | x (x) |
| | ICF not signed prior to study procedures | x (x) | x (x) | x (x) | x (x) |
| | Other | x (x) | x (x) | x (x) | x (x) |
| Treatment administration schedule | Any type | x (x) | x (x) | Placebo (N=X) | x (x) |
| | Out of window visit | x (x) | x (x) | x (x) | x (x) |
| | Missed visit/visit not conducted | x (x) | x (x) | x (x) | x (x) |
| | Missed treatment administration | x (x) | x (x) | x (x) | x (x) |
| | Delayed treatment administration | x (x) | x (x) | x (x) | x (x) |
| | Other | x (x) | x (x) | x (x) | x (x) |
| Follow-up visit schedule | Any type | x (x) | x (x) | x (x) | x (x) |
| • | Out of window visit | x (x) | x (x) | x (x) | x (x) |
| | Missed visit/visit not conducted | x (x) | x (x) | x (x) | x (x) |
| | Other | x (x) x (x) x (x) | x (x) | x (x) | |
| Protocol procedure/assessment | Any type | x (x) | x (x) | x (x) | x (x |
| | Incorrect version of ICF signed | x (x) | x (x) | x (x) | x (x) |
| | Blood not collected | x (x) | x (x) | x (x) | x (x) |
| | Urine not collected | x (x) | x (x) | x (x) | x (x) |
| | Other specimen not collected | x (x) | x (x) | x (x) | x (x) |
| | Too few aliquots obtained | x (x) | x (x) | x (x) | x (x) |
| | Specimen result not obtained | x (x) | x (x) | x (x) | x (x) |
| | Required procedure not conducted | x (x) | x (x) | x (x) | x (x) |
| | Required procedure done incorrectly | x (x) | x (x) | x (x) | x (x) |
| | Study product temperature excursion | x (x) | x (x) | x (x) | x (x) |
| | Specimen temperature excursion | x (x) | x (x) | | x (x) |
| | Other | x (x) | x (x) | x (x) | x (x) |
| Treatment administration | Any type | x (x) | x (x) | | x (x) |
| | Required procedure done incorrectly | x (x) | x (x) | | x (x) |
| | Study product temperature excursion | x (x) | x (x) | | x (x) |
| | Other | x (x) | x (x) | x (x) | x (x) |
| Blinding policy/procedure | Any type | x (x) | x (x) | x (x) | x (x) |
| | Treatment unblinded | x (x) | x (x) | x (x) | x (x) |
| | Other | x (x) | x (x) | x (x) | x (x) |
| Note: N = Number of subjects in Sa | | | | | |

# 14.1 Description of Study Subjects

# 14.1.1 Disposition of Subjects

**Table 2:** Subject Disposition by Dose Group

| | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| <b>Subject Disposition</b> | n (%) | n (%) | n (%) | n (%) |
| Screened | - | - | - | x (-) |
| Enrolled/Randomized | x (100) | x (100) | x (100) | x (100) |
| Received Study Product | x (x) | x (x) | x (x) | x (x) |
| Completed all PK Blood Draws | x (x) | x (x) | x (x) | x (x) |
| Completed Final Study Visit | x (x) | x (x) | x (x) | x (x) |
| Early Termination | x (x) | x (x) | x (x) | x (x) |
| Note: N= Number of subjects randomized. | l | ı | | I |

# **Table 3:** Analysis Populations by Dose Group

[Implementation Note: Although subjects may meet multiple criteria for exclusion, they will be counted under only one reason for exclusion in this table. Priority for assigning reasons for exclusions will follow the order in the table.]

| | | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) | All<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|
| <b>Analysis Populations</b> | Reason Subjects Excluded | n (%) | n (%) | n (%) | n (%) |
| Safety Population | No study product received | x (x) | x (x) | x (x) | x (x) |
| PK Analysis Population | Any Reason | x (x) | x (x) | x (x) | x (x) |
| | Subject received placebo or was enrolled in Cohort 1 | x (x) | x (x) | x (x) | x (x) |
| | Assigned dose not received or completed | x (x) | x (x) | x (x) | x (x) |
| | Subject has no measurable concentration of drug | x (x) | x (x) | x (x) | x (x) |
| PK Analysis Subset | Any Reason | x (x) | x (x) | x (x) | x (x) |
| | Exclusion from PK Analysis Population | x (x) | x (x) | x (x) | x (x) |
| | Has protocol deviations that potentially impact PK | x (x) | x (x) | x (x) | x (x) |
| | PK data insufficient to estimate any PK parameters | x (x) | x (x) | x (x) | x (x) |
| Note: N= Number of subject | ets randomized. | • | 1 | | |

### **Table 4:** Ineligibility Summary of Screen Failures

[Implementation Note: Criteria displayed in the actual table will copy verbatim from the protocol with appropriate footnotes. The final summary table will include only inclusion/exclusion criterion with at least 1 subject. Criteria that were not met by any subjects will be excluded from final table.]

| | | Subjects | Excluded |
|---|---|---|---|
| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | % b |
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | х | 100 |
| Inclusion | Any inclusion criterion | X | x |
| | Willing and able to provide written informed consent and authorization for use of PHI | x | x |
| | Willing and able to comply with protocol requirements and is likely to complete the study as planned | x | x |
| | Males are vasectomized or agree to use barrier contraception from first dose through 18 weeks post last dose of IP | X | x |
| | Females are of non-childbearing potential or agree to use specified BC for 30 days pre and post-dose | X | x |
| | Subject is in good health as deemed by the Investigator | X | x |
| | Subject has a BMI between 18.5 and 35.0 kg/m <sup>2</sup> , inclusive and a minimum weight of 50 kg | х | x |
| | Subject must refrain from strenuous physical activity from screening until completion of the trial | X | x |
| | Subjects must refrain from OTC/Rx meds, nutrition supplements from 14 days pre-dose to final visit | X | x |
| | Subject has adequate venous access for blood collection | X | x |
| Exclusion | Any exclusion criterion | x | x |
| | Subjects with clinical laboratory values outside the site reference ranges prior to initial dosing | x | x |
| | Abnormal ECGs. | X | x |
| | Female subject is pregnant, lactating or planning to become pregnant | X | x |
| | Received any prescription medications (with exceptions) within 14 days before first dose | Х | x |
| | Received any non-prescription medications, vitamins or supplements within 14 days of initial dose | X | x |
| | Current smoker or tobacco use within 90 days prior to dosing or while subject is enrolled in study | X | x |
| | History of illicit/illegal drug use, alcohol/substance abuse, or vaping of non-nicotine products | X | x |
| | Consumed alcohol <= 48 hours of xanthines/caffeine <= 24 hours before first dose until discharge | X | x |
| | Received any live or killed vaccines or immunoglobulins within 14 days of dosing | X | x |
| | Donated blood or blood products or experienced significant blood loss within 60 days of dosing | X | x |
| | Received a blood transfusion within 14 days of dosing | х | х |

| | | Subjects Exclude | |
|---|---|---|---|
| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | nª | % b |
| | Previous participation in any trial within 28 days of dosing or plans to enroll in another trial | х | x |
| | The PI considers that the subject should not participate in the trial | х | x |
| Eligible but Not Enrolled | Any Reason | X | x |
| | [Reason 1] | x | x |
| | [Reason 2] | x | x |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.
<sup>b</sup> Denominator for percentages is the total number of screen failures.

# 14.1.2 Demographic Data by Dose Group

Table 5: Summary of Categorical Demographic and Baseline Characteristics by Dose Group

| | | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| Variable | Characteristic | n (%) | n (%) | n (%) | n (%) |
| Sex | Male | x (x) | x (x) | x (x) | x (x) |
| | Female | x (x) | x (x) | x (x) | x (x) |
| Ethnicity | Not Hispanic or Latino | x (x) | x (x) | x (x) | x (x) |
| | Hispanic or Latino | x (x) | x (x) | x (x) | x (x) |
| | Not Reported | x (x) | x (x) | x (x) | x (x) |
| | Unknown | x (x) | x (x) | x (x) | x (x) |
| Race | American Indian or Alaska Native | x (x) | x (x) | x (x) | x (x) |
| | Asian | x (x) | x (x) | x (x) | x (x) |
| | Native Hawaiian or Other Pacific Islander | x (x) | x (x) | x (x) | x (x) |
| | Black or African American | x (x) | x (x) | x (x) | x (x) |
| | White | x (x) | x (x) | x (x) | x (x) |
| | Multi-Racial | x (x) | x (x) | x (x) | x (x) |
| | Unknown | x (x) | x (x) | x (x) | x (x) |
| Note: N= Number of | f subjects randomized. | 1 | • | | 1 |
Table 6: Summary of Continuous Demographic and Baseline Characteristics by Dose Group

| Variable | Statistic | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| Age (years) | Mean | х | х | x | х |
| | SD | х | х | x | х |
| | Median | х | х | x | х |
| | Min | X | х | x | х |
| | Max | X | х | x | х |
| Height (cm) | Mean | X | х | x | х |
| | SD | X | х | x | х |
| | Median | х | х | x | х |
| | Min | X | х | x | х |
| | Max | х | х | x | х |
| Weight (kg) | Mean | х | х | x | х |
| | SD | х | х | x | х |
| | Median | х | х | x | х |
| | Min | X | x | x | x |
| | Max | X | x | x | x |
| BMI (kg/m²) | Mean | X | x | x | x |
| | SD | х | x | x | х |
| | Median | х | x | x | х |
| | Min | х | x | x | х |
| | Max | X | х | х | X |

#### 14.1.3 Prior and Concurrent Medical Conditions

Table 7: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Dose Group

| | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| MedDRA System Organ Class | n (%) | n (%) | n (%) | n (%) |
| Any SOC | | | | |
| [SOC 1] | | | | |
| [SOC 2] | | | | |
| Note: N= Number of subjects randomized. | | | | |

### 14.3 Safety Data

#### 14.3.1 Displays of Adverse Events

## **Table 8:** Overall Summary of Adverse Events by Dose Group

[Implementation Note: Abnormal laboratory AEs assessed using the protocol toxicity tables will not be included in this summary.]

| | SAD<br>Any Dose<br>(N=X) | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) |
|---|---|---|---|---|
| Subjects with | n (%) | n (%) | n (%) | n (%) |
| At least one solicited reactogenicity event | x (x) | x (x) | x (x) | x (x) |
| At least one ulceration | x (x) | x (x) | x (x) | x (x) |
| At least one mild (or worse) solicited reactogenicity event | x (x) | x (x) | x (x) | x (x) |
| At least one moderate (or worse) solicited reactogenicity event | x (x) | x (x) | x (x) | x (x) |
| At least one severe solicited reactogenicity event | x (x) | x (x) | x (x) | x (x) |
| At least one adverse event | x (x) | x (x) | x (x) | x (x) |
| At least one related adverse event | x (x) | x (x) | x (x) | x (x) |
| At least one mild (or worse) related adverse event | x (x) | x (x) | x (x) | x (x) |
| At least one moderate (or worse) related adverse event | x (x) | x (x) | x (x) | x (x) |
| At least one severe related adverse event | x (x) | x (x) | x (x) | x (x) |
| At least one serious adverse event | x (x) | x (x) | x (x) | x (x) |
| At least one related, serious adverse event | x (x) | x (x) | x (x) | x (x) |
| At least one adverse event leading to early termination | x (x) | x (x) | x (x) | x (x) |
| Note: N = Number of subjects in Safety Population | <b>.</b> | 1 | ı | 1 |

#### **14.3.1.1** Solicited Reactogenicity Events

# Table 9: Number and Percentage of Subjects Experiencing Solicited Reactogenicity Symptoms with 95% Confidence Intervals by Symptom and Dose Group

[Implementation Note: Each subject is counted once per symptom.]

| | SAD<br>Any Dose<br>(N=X) | | SAD<br>1 mg<br>(N=X) | | | SAD<br>10 mg<br>(N=X) | | | Placebo<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | X | xx | x.x, x.x | X | XX | x.x, x.x | X | xx | x.x, x.x | X | xx | x.x, x.x |
| Pain | | | | | | | | | | | | |
| Tenderness | | | | | | | | | | | | |
| Pruritus (Itching) | | | | | | | | | | | | |
| Ecchymosis (Bruising), Functional Grade | | | | | | | | | | | | |
| Ecchymosis (Bruising), Measurement Grade | | | | | | | | | | | | |
| Induration (Hardness)/ Swelling, Functional Grade | | | | | | | | | | | | |
| Induration (Hardness)/ Swelling, Measurement<br>Grade | | | | | | | | | | | | |
| Erythema (Redness), Functional Grade | | | | | | | | | | | | |
| Erythema (Redness), Measurement Grade | | | | | | | | | | | | |
| Nodule, Functional Grade | | | | | | | | | | | | |
| Nodule, Measurement Grade | | | | | | | | | | | | |
| Ulceration, Functional Grade | | | | | | | | | | | | |
| Ulceration, Measurement Grade | | | | | | | | | | | | |
| Note: N = Number of subjects in the Safety Populati | on. | | • | | | • | • | | • | | • | - |

Table 10: Number and Percentage of Subjects Experiencing Solicited Reactogenicity Symptoms with 95% Confidence Intervals by Symptom, Severity, and Dose Group

[Implementation Note: Each subject is counted once per symptom.]

| | | | SAD<br>Any Dose<br>(N=X) | | SAD<br>1 mg<br>(N=X) | | SAD<br>10 mg<br>(N=X) | | | Placebo<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | None | X | XX | x.x, x.x | Х | XX | x.x, x.x | Х | XX | x.x, x.x | Х | XX | x.x, x.x |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Tenderness | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Pruritus (Itching) | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Ecchymosis (Bruising), Functional Grade | None | | | | | | | | | | | | |
| Ecchymosis (Bruising), Measurement Grade | None | | | | | | | | | | | | |
| Induration (Hardness)/ Swelling, Functional Grade | | | | | | | | | | | | | |

| | | SAD<br>Any Dose<br>(N=X) | | SAD<br>1 mg<br>(N=X) | | SAD<br>10 mg<br>(N=X) | | Placebo<br>(N=X) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Induration (Hardness)/ Swelling, Measurement Grade | | | | | | | | | | | | | |
| Erythema (Redness), Functional Grade | | | | | | | | | | | | | |
| Erythema (Redness), Measurement Grade | | | | | | | | | | | | | |
| Nodule, Functional Grade | | | | | | | | | | | | | |
| Nodule, Measurement Grade | | | | | | | | | | | | | |
| Ulceration, Functional Grade | | | | | | | | | | | | | |
| Ulceration, Measurement Grade | | | | | | | | | | | | | |
| Note: N = Number of subjects in Safety Population | | | | | | | | | | | | | |

Table 11: Number and Percentage of Subjects Experiencing Solicited Reactogenicity Symptoms by Symptom, Severity, Time Point, and Dose Group

| | | | N | one | Mi | ld | Mod | erate | Se | vere |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose Group | Time Point | N | n | % | n | % | n | % | n | % |
| Any Symptoms | | | | | | | | | | |
| SAD Any Dose | Max Severity Post Baseline | | | | | | | | | |
| | Day 1, 1 h Post-Dose | | | | | | | | | |
| | Day 1, 4 h Post-Dose | | | | | | | | | |
| | Day 2 | | | | | | | | | |
| | Day 3 | | | | | | | | | |
| | Day 4 | | | | | | | | | |
| | Day 5 | | | | | | | | | |
| | Day 6 | | | | | | | | | |
| | Day 7 | | | | | | | | | |
| | Max Severity Day 8 to Day 14 | | | | | | | | | |
| | Max Severity Day 15 to Day 21 | | | | | | | | | |
| | Max Severity Day 22 to Final Visit | | | | | | | | | |
| SAD 1 mg | Max Severity Post Baseline | | | | | | | | | |
| SAD 10 mg | Max Severity Post Baseline | | | | | | | | | |
| Placebo | Max Severity Post Baseline | | | | | | | | | |
| Pain | | | | | | | | | | |
| SAD Any Dose | | | | | | | | | | |
| SAD 1 mg | | | | | | | | | | |
| SAD 10 mg | | | | | | | | | | |
| Tenderness | | | | | | | | | | |
| Ecchymosis (Bru | nising), Functional Grade | | | | | | | | | |
| Ecchymosis (Bru | nising), Measurement Grade | | | | | | | | | |
| Induration (Har | dness)/ Swelling, Functional Grade | | | | | | | | | |
| Induration (Har | dness)/ Swelling, Measurement Grade | e | | | | | | | | |
| Erythema (Redn | ess), Functional Grade | | | | | | | | | |
| Erythema (Redn | ess), Measurement Grade | | | | | | | | | |
| Nodule, Function | nal Grade | | | | | | | | | |
| Nodule, Measure | ement Grade | | | | | | | | | |
| Ulceration, Func | tional Grade | | | | | | | | | |
| Ulceration, Meas | surement Grade | | | | | | | | | |
| Note: $N = Numl$ | ber of subjects in Safety Population | with so | licited re | eactogeni | city sympto | oms asses | ssed at th | ne respec | tive time | point. |

#### 14.3.1.2 Unsolicited Adverse Events

# Table 12: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Dose Group

[Implementation Note: If there is only 1 PT for an SOC, there will be no "Any PT" row.]

| Dose Group | MedDRA System Organ<br>Class | MedDRA Preferred<br>Term | N | n (%) | 95% CI | Number of<br>Events |
|---|---|---|---|---|---|---|
| SAD Any Dose | Any SOC | Any PT | x | x (x) | (x.x, x.x) | X |
| | [SOC 1] | Any PT | x | x (x) | (x.x, x.x) | X |
| | | [PT 1] | х | x (x) | (x.x, x.x) | X |
| | | [PT 2] | x | x (x) | (x.x, x.x) | X |
| | Any SOC | Any PT | x | x (x) | (x.x, x.x) | X |
| SAD 1 mg | | | | | | |
| Note: N = Number of s | subjects in Safety Population | • | • | | • | • |

Table 13: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship, and Dose Group

[Implementation Note: If there is only 1 PT for an SOC, there will be no "Any PT" row.]

| Dose Group | MedDRA System Organ<br>Class | MedDRA Preferred<br>Term | Severity | N | Related n(%) | Not Related<br>n (%) | Total<br>n (%) |
|---|---|---|---|---|---|---|---|
| SAD Any Dose | Any SOC | Any PT | Any Severity | х | x (x) | x (x) | x (x) |
| | | | Mild | х | x (x) | x (x) | x (x) |
| | | | Moderate | х | x (x) | x (x) | x (x) |
| | | | Severe | х | x (x) | x (x) | x (x) |
| | [SOC 1] | Any PT | Any Severity | х | x (x) | x (x) | x (x) |
| | | | Mild | х | x (x) | x (x) | x (x) |
| | | | Moderate | х | x (x) | x (x) | x (x) |
| | | | Severe | х | x (x) | x (x) | x (x) |
| | | [PT 1] | Any Severity | х | x (x) | x (x) | x (x) |
| | | | Mild | х | x (x) | x (x) | x (x) |
| | | | Moderate | х | x (x) | x (x) | x (x) |
| | | | Severe | х | x (x) | x (x) | x (x) |
| | | | | х | x (x) | x (x) | x (x) |
| SAD 1 mg | Any SOC | Any PT | Any Severity | х | x (x) | x (x) | x (x) |
| Note: N = Number | r of subjects in Safety Population | on | • | • | • | | |

#### 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

#### **Table 14:** Listing of Serious Adverse Events

[Implementation Note: This listing is included in the table shells document, as it is included in the body of the abbreviated CSR. If the event is ongoing (no stop date), indicate "ongoing" for the "Duration". If more than one reason is selected for the reason reported as an SAE, list all reasons in the column, separated by a comma. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon. Listing should be sorted by Dose Group, Subject ID, and AE Number.]

| Adverse<br>Event | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term | Study Day | Duration of<br>AE in Days | Study Day the<br>Event Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship to<br>Study Treatment<br>(Alternate Etiology) | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose Gro | up: , Subject ID: | , AE Number: | | | | | | | | | |
| Comments | s: | | | | | | | | | | |
| Dose Gro | up: , Subject ID: | , AE Number: | | | | | | | | | |
| Comment | s: | | | | | | | | • | | |

#### Table 15: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

[Implementation Note: This listing is included in the tables document, as it is included in the body of the abbreviated CSR. If the event is ongoing (no stop date), indicate "ongoing" in the "Duration" column. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon. Listing should be sorted by Dose Group, Subject ID, and AE Number.]

| Adverse<br>Event | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred Term | Study Day | Duration of<br>AE in Days | Severity | Relationship to<br>Study Treatment<br>(Alternate Etiology) | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| Dose Group: , S | Subject ID: , AE N | umber: | | | | | | | |
| Comments: | | | | | | | | | |
| Dose Group: , S | Subject ID: , AE Ni | umber: | | | | | | | |
| Comments: | | | | | | | | | |

### 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

#### 14.3.4 Abnormal Laboratory Value Listings (by Subject)

#### **Table 16:** Listing of Abnormal Laboratory Results – Chemistry

[Implementation Note: This listing is included in the table shells document, as it is included in the body of the abbreviated CSR. This listing includes all abnormal Chemistry results (laboratory results outside of the normal range defined in the protocol). Normal chemistry results for other parameters that occurred on the same visit as the abnormal result will not be listed. There is a separate, complete listing of all Chemistry results. In the Laboratory Parameter column, indicate the units (LB.LBSTRESU) after the parameter, e.g., Sodium (mEq/L). This listing is not color-coded. Results that are outside the normal range but not mild, moderate, or severe will have ONR listed as severity. Similarly, results that meet grading criteria of mild, moderate, or severe but which are not treatment emergent (not worse than baseline) will be shown as ONR.

| Dose Group | Subject ID | Sex | Time Point | Date of<br>Assessment | Laboratory Parameter (Units) | Result | Severity |
|---|---|---|---|---|---|---|---|

#### Table 17: Listing of Abnormal Laboratory Results - Hematology

[Implementation Note: This listing is included in the table shells document, as it is included in the body of the abbreviated CSR. This listing includes all abnormal Hematology results (laboratory results outside of the normal range defined in the protocol). Normal hematology results for other parameters that occurred on the same visit as the abnormal result will not be listed. There is a separate, complete listing of all Hematology results. In the Laboratory Parameter column, indicate the units (LB.LBSTRESU) after the parameter, e.g., Hemoglobin (g/dL). This listing is not color-coded. Results that are outside the normal range but not mild, moderate, or severe will have ONR listed as severity. Similarly, results that meet grading criteria of mild, moderate, or severe but which are not treatment emergent (not worse than baseline) will be shown as ONR..

| Dose Group | Subject ID | Sex | Time Point | Date of<br>Assessment | Laboratory Parameter (Units) | Result | Severity |
|---|---|---|---|---|---|---|---|

#### **Table 18:** Listing of Abnormal Laboratory Results - Coagulation

[Implementation Note: This listing is included in the table shells document, as it is included in the body of the abbreviated CSR. This listing includes all abnormal Coagulation results (laboratory results outside of the normal range defined in the protocol). Normal coagulation results for other parameters that occurred on the same visit as the abnormal result will not be listed. There is a separate, complete listing of all Coagulation results. In the Laboratory Parameter column, indicate the units (LB.LBSTRESU) after the parameter, e.g., (seconds). This listing is not color-coded. Results that are outside the normal range but not mild, moderate, or severe will have ONR listed as severity. Similarly, results that meet grading criteria of mild, moderate, or severe but which are not treatment emergent (not worse than baseline) will be shown as ONR.

| Dose Group | Subject ID | Time Point | Date of<br>Assessment | Laboratory Parameter (Units) | Result | Severity |
|---|---|---|---|---|---|---|

#### **Table 19:** Listing of Abnormal Laboratory Results - Urinalysis

[Implementation Note: This listing is included in the table shells document, as it is included in the body of the abbreviated CSR. This listing includes all abnormal Urinalysis results (laboratory results outside of the normal range defined in the protocol). Normal urinalysis results for other parameters that occurred on the same visit as the abnormal result will not be listed. There is a separate, complete listing of all Urinalysis results. In the Laboratory Parameter column, indicate the units (LB.LBSTRESU) after the parameter, e.g., Leukocytes by Microscopy (/hpf). This listing is not color-coded. Results that are outside the normal range but not mild, moderate, or severe will have ONR listed as severity. Similarly, results that meet grading criteria of mild, moderate, or severe but which are not treatment emergent (not worse than baseline) will be shown as ONR.

| Dose Group | Subject ID | Sex | Time Point | Date of<br>Assessment | Laboratory Parameter (Units) | Result | Severity |
|---|---|---|---|---|---|---|---|
| | | | | | Occult Blood by Dipstick | Negative | |

#### 14.3.5 Displays of Laboratory Results

#### 14.3.5.1 Chemistry Results

### Table 20: Chemistry Toxicity Grade by Parameter, Severity, Dose Group, and Time Point

[Implementation Note: Severity will be graded based on toxicity criteria in protocol. If there is not at least 1 Mild, Moderate, or Severe Event for Max Severity Post-Baseline, then only the Max Severity Post-Baseline row will be shown for the parameter. Toxicities representing an increase in the laboratory result will be summarized separately from decreases.]

| | | | Mild | Moderate | Severe |
|---|---|---|---|---|---|
| Dose Group | Time Point | N | n (%) | n (%) | n (%) |
| Any Parameter | | | | | |
| SAD Any Dose | Baseline | X | x (x) | x (x) | x (x) |
| | Max Severity Post-Baseline | x | x (x) | x (x) | x (x) |
| | Day 2 | X | x (x) | x (x) | x (x) |
| | Day 7 | X | x (x) | x (x) | x (x) |
| | Final Visit | X | x (x) | x (x) | x (x) |
| SAD 1 mg | Baseline | X | x (x) | x (x) | x (x) |
| | | X | x (x) | x (x) | x (x) |
| SAD 10 mg | Baseline | x | x (x) | x (x) | x (x) |
| | | X | x (x) | x (x) | x (x) |
| Placebo | Baseline | X | x (x) | x (x) | x (x) |
| | | X | x (x) | x (x) | x (x) |
| Sodium, Decrease | | | | | |
| SAD Any Dose | Baseline | X | x (x) | x (x) | x (x) |
| ••• | | X | x (x) | x (x) | x (x) |

Notes: The "Max Severity Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

N=Number of subjects in the Safety Population with the laboratory result assessed at the respective time point.

Table 21: Chemistry Change from Baseline by Parameter, Dose Group, and Time Point

| | | | | Change fr | om Baseline | |
|---|---|---|---|---|---|---|
| Dose Group | Time Point | N | Mean | SD | Median | Min, Max |
| Sodium (mEq/L) | <u>.</u> | | | | | |
| SAD Any Dose | Day 2 | х | Х | Х | Х | x, x |
| | Day 7 | х | Х | Х | X | x, x |
| | Final Visit | х | Х | Х | X | x, x |
| SAD 1 mg | Day 2 | х | | | | |
| | | х | Х | Х | X | x, x |
| SAD 10 mg | Day 2 | х | | | | |
| | | х | Х | X | X | x, x |
| | | х | Х | X | X | x, x |
| Placebo | Day 2 | х | Х | Х | Х | x, x |
| | | х | Х | Х | Х | x, x |
| Potassium (mEq/L) | · | | | | | |
| SAD Any Dose | Day 2 | х | Х | Х | Х | x, x |
| | | Х | Х | Х | X | x, x |

#### 14.3.5.2 Hematology Results

#### Table 22: Hematology Toxicity Grade by Parameter, Severity, Dose Group, and Time Point

[Implementation Note: Severity will be graded based on toxicity criteria in protocol. If there is not at least 1 Mild, Moderate, or Severe Event for Max Severity Post-Baseline, then only the Max Severity Post-Baseline row will be shown for the parameter. Toxicities representing an increase in the laboratory result will be summarized separately from decreases.]

This table will repeat Table 20 for Hematology parameters.

#### Table 23: Hematology Change from Baseline by Parameter, Dose Group, and Time Point

This table will repeat Table 21 for Hematology parameters.

#### 14.3.5.3 Coagulation Clinical Laboratory Results

#### Table 24: Coagulation Toxicity Grade by Parameter, Dose Group, and Time Point

[Implementation Note: Severity will be graded based on toxicity criteria in protocol. If there is not at least 1 Mild, Moderate, or Severe Event for Max Severity Post-Baseline, then only the Max Severity Post-Baseline row will be shown for the parameter. Toxicities representing an increase in the laboratory result will be summarized separately from decreases.]

This table will repeat Table 20 for Coagulation parameters.

#### Table 25: Coagulation Change from Baseline by Parameter, Dose Group, and Time Point

This table will repeat Table 21 for Coagulation parameters.

#### 14.3.5.4 Urinalysis Results

#### Table 26: Urinalysis Toxicity Grade by Parameter, Severity, Dose Group, and Time Point

[Implementation Note: Severity will be graded based on toxicity criteria in protocol. If there is not at least 1 Mild, Moderate, or Severe Event for Max Severity Post-Baseline, then only the Max Severity Post-Baseline row will be shown for the parameter. Toxicities representing an increase in the laboratory result will be summarized separately from decreases.]

This table will repeat Table 20 for Urinalysis parameters.

## 14.3.6 Displays of Vital Signs

Table 27: Vital Sign Toxicity Grade by Parameter, Severity, Dose Group, and Time Point

[Implementation Note: If there is not at least 1 Mild, Moderate, or Severe Event for Max Severity Post-Baseline, then only the Max Severity Post-Baseline row will be shown for the parameter.]

| Dose Group | Time Point | N | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) |
|---|---|---|---|---|---|
| Any Parameter | | | | , | |
| SAD Any Dose | Baseline | х | x (x) | x (x) | x (x) |
| | Max Severity Post Baseline | | | | |
| | Day 1, 15 minutes Post-Dose | х | x (x) | x (x) | x (x) |
| | Day 1, 1 h Post-Dose | х | x (x) | x (x) | x (x) |
| | Day 1, 2 h Post-Dose | х | x (x) | x (x) | x (x) |
| | Day 2 | х | x (x) | x (x) | x (x) |
| | Day 4 | х | x (x) | x (x) | x (x) |
| | Day 7 | х | x (x) | x (x) | x (x) |
| | Day 14 | х | x (x) | x (x) | x (x) |
| | Final Visit | х | x (x) | x (x) | x (x) |
| SAD 1 mg | Baseline | х | x (x) | x (x) | x (x) |
| | | х | x (x) | x (x) | x (x) |
| SAD 10 mg | Baseline | х | x (x) | x (x) | x (x) |
| | | х | x (x) | x (x) | x (x) |
| Placebo | Baseline | х | x (x) | x (x) | x (x) |
| | | х | x (x) | x (x) | x (x) |
| Systolic Blood Pressu | re, Decrease | | | , | |
| SAD Any Dose | Baseline | х | x (x) | x (x) | x (x) |
| | | х | x (x) | x (x) | x (x) |

Notes: The "Max Severity Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

N = Number of subjects in Safety Population with the vital sign assessed for the respective time point.

Table 28: Vital Sign Change from Baseline by Parameter, Dose Group, and Time Point

| | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|
| Dose Group | Time Point | N | Mean | SD | Median | Min, Max |
| Systolic Blood Pressure | (mmHg) | | | | | |
| SAD Any Dose | Day 1, 15 minutes Post-Dose | х | х | Х | х | x, x |
| | Day 1, 1 h Post-Dose | х | х | Х | х | x, x |
| | Day 1, 2 h Post-Dose | х | X | Х | х | x, x |
| | Day 2 | х | X | Х | х | x, x |
| | Day 4 | х | X | Х | х | x, x |
| | Day 7 | X | Х | X | Х | x, x |
| | Day 14 | X | X | X | х | x, x |
| | Final Visit | X | X | X | х | x, x |
| SAD 1 mg | Day 1, 15 minutes Post-Dose | х | X | Х | х | x, x |
| | | х | X | Х | х | x, x |
| SAD 10 mg | Day 1, 15 minutes Post-Dose | х | X | Х | х | x, x |
| | | х | X | Х | х | x, x |
| Placebo | Day 1, 30 minutes Post-Dose | х | X | Х | х | x, x |
| | | | X | X | х | x, x |
| Diastolic Blood Pressur | re (mmHg) | | | | | |
| SAD Any Dose | Day 1, 15 minutes Post-Dose | x | х | х | х | x, x |
| | | X | х | X | Х | x, x |
| Note: N=Number of sub | jects in the Safety Population with the la | boratory resu | It assessed at the | respective time p | oint. | 1 |

#### 14.3.7 Displays of ECG Measurements

Table 29: ECG Overall Interpretations, Post Dose Compared to Baseline by Dose Group and Time Point

| ECG Interpretation | SAD Any Dose<br>n (%) | SAD 1 mg<br>n (%) | SAD 10 mg<br>n (%) | Placebo<br>n (%) |
|---|---|---|---|---|
| Day 1, 4 h Post-Dose | | | | |
| N | x | Х | x | X |
| Normal at Both Times | x (x) | x (x) | x (x) | x (x) |
| Normal to Abnormal, NCS | x (x) | x (x) | x (x) | x (x) |
| Normal to Abnormal, CS | | | | |
| Abnormal, NCS at Both Times | x (x) | x (x) | x (x) | x (x) |
| Abnormal, NCS to Abnormal, CS | | | | |
| Abnormal, NCS to Normal | x (x) | x (x) | x (x) | x (x) |
| Day 7 | | | | |
| N | х | x | x | X |
| Normal at Both Times | x (x) | x (x) | x (x) | x (x) |
| | x (x) | x (x) | x (x) | x (x) |
| Final Visit | | | | |
| N | x | x | x | X |
| Normal at Both Times | x (x) | x (x) | x (x) | x (x) |
| | x (x) | x (x) | x (x) | x (x) |

Notes: N = Number of subjects in Safety Population with the ECG results assessed at the respective time point. CS= clinically significant; NCS= not clinically significant.

#### Table 30: ECG Toxicity Grade by Parameter, Severity, Dose Group, and Time Point

[Implementation Note: If there is not at least 1 Mild, Moderate, or Severe Event for Max Severity Post-Baseline, then only the Max Severity Post-Baseline row will be shown for the parameter.]

| Dose Group | Time Point | N | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) |
|---|---|---|---|---|---|
| PR Interval | | | | | |
| SAD Any Dose | Baseline | х | x (x) | x (x) | x (x) |
| | Max Severity Post Baseline | | | | |
| | Day 1, 4 h Post-Dose | х | x (x) | x (x) | x (x) |
| | Day 7 | х | x (x) | x (x) | x (x) |
| | Final Visit | х | x (x) | x (x) | x (x) |
| SAD 1 mg | Baseline | х | x (x) | x (x) | x (x) |
| | | х | x (x) | x (x) | x (x) |
| SAD 10 mg | Baseline | х | x (x) | x (x) | x (x) |
| | | х | x (x) | x (x) | x (x) |
| Placebo | Baseline | х | x (x) | x (x) | x (x) |
| | | х | x (x) | x (x) | x (x) |
| QTcF Interval | | | | | |
| SAD Any Dose | Baseline | х | x (x) | x (x) | x (x) |
| | | х | x (x) | x (x) | x (x) |

Notes: The "Max Severity Post Baseline" rows indicate the maximum severity of ECG Results Related to study treatment experienced by each subject at any time point post baseline, including unscheduled assessments.

N = Number of subjects in Safety Population with the ECG results assessed at the respective time point.

Table 31: ECG Change from Baseline by Parameter, Dose Group, and Time Point

| | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|
| Dose Group | Time Point | N | Mean | SD | Median | Min, Max |
| PR Interval (msec) | | | | | | |
| SAD Any Dose | Day 1, 4 h Post-Dose | X | х | х | Х | х, х |
| | Day 7 | х | х | х | Х | x, x |
| | Final Visit | х | х | х | Х | х, х |
| SAD 1 mg | Day 1, 4 h Post-Dose | х | х | х | х | х, х |
| | | х | х | х | х | x, x |
| SAD 10 mg | Day 1, 4 h Post-Dose | х | Х | х | х | x, x |
| | | х | Х | х | х | x, x |
| Placebo | Day 1, 4 h Post-Dose | х | Х | х | х | x, x |
| | | х | Х | х | х | x, x |
| QRS Duration (msec) | | | | | | |
| SAD Any Dose | Day 1, 4 h Post-Dose | X | х | х | Х | x, x |
| | | x | х | х | X | x, x |
| Note: $N = Number of s$ | subjects in Safety Population with the | ECG results as | sessed at the resp | pective time point. | 1 | • |

#### Table 32: Summary of QTcF by Dose Group and Time Point

[Implementation Note: For all QTcF categories that specified gender, N based on gender should be used for calculating proportions]

| | | SAD Any Dose | SAD 1 mg | SAD 10 mg | Placebo |
|---|---|---|---|---|---|
| QTcF Category | Time Point | n / N (%) | n / N (%) | n / N (%) | n / N (%) |
| QTcF >450 ms, Male | Day 1, 4 h Post-Dose | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| | Day 7 | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| | Final Visit | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| QTcF >470 ms, Female | Day 1, 4 h Post-Dose | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| | | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| QTcF >480 ms | Day 1, 4 h Post-Dose | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| | | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| QTcF >500 ms | Day 1, 4 h Post-Dose | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| | | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| 30 ms ≤ QTcF increases from baseline < 60 ms | Day 1, 4 h Post-Dose | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| | | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| QTcF increases from baseline ≥ 60 ms | Day 1, 4 h Post-Dose | x / x (x) | x / x (x) | x / x (x) | x / x (x) |
| | | x / x (x) | x / x (x) | x / x (x) | x / x (x) |

N= Number of subjects in Safety Population with the ECG results assessed at the respective time point. N is calculated based on specified sex for "QTcF >450 ms, Male" and "QTcF >470 ms, Female" categories.

#### 14.4 Summary of Concomitant Medications

# Table 33: Number and Percentage of Subjects with Prior Medications by WHO Drug Classification and Dose Group

[Implementation Note: Include prior medications (medications with an end date prior to first dose) only.]

| WHO Drug Code | WHO Drug Code | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| Level 1, Anatomic Group | Level 2, Therapeutic Subgroup | n (%) | n (%) | n (%) | n (%) |
| Any Level 1 Codes | Any Level 2 Codes | | | | |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | |
| | [ATC 2 - 1] | | | | |
| | [ATC 2 - 2] | | | | |
| | [ATC 2 - 3] | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | |
| | [ATC 2 - 2] | | | | |
| | [ATC 2 - 3] | | | | |
| Note: $N = Number of subjects in S$ | Safety Population | | • | | • |

# Table 34: Number and Percentage of Subjects with Concomitant Medications by WHO Drug Classification and Dose Group

[Implementation Note: Include concomitant medications (medications that are ongoing or that have an end date after first dose) only]

| WHO Drug Code | WHO Drug Code | SAD<br>1 mg<br>(N=X) | SAD<br>10 mg<br>(N=X) | Placebo<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| Level 1, Anatomic Group | Level 2, Therapeutic Subgroup | n (%) | n (%) | n (%) | n (%) |
| Any Level 1 Codes | Any Level 2 Codes | | | | |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | |
| | [ATC 2 - 1] | | | | |
| | [ATC 2 - 2] | | | | |
| | [ATC 2 - 3] | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | |
| | [ATC 2 - 2] | | | | |
| | [ATC 2 - 3] | | | | |
| Note: $N = Number of subjects in S$ | Safety Population | | • | • | • |

#### 14.5 Pharmacokinetics

Table 35: Rezafungin Concentrations in Plasma, SAD 10 mg Dose Group

| | Nominal Time <sup>a</sup> (h) | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | 0 | 0.5 | 1 | 2 | 4 | 6 | 8 | 12 | 24 | 48 | 96 | 144 | 312<br>(Day 14) | 696<br>(Day 30) |
| PHU.00123 | х | х | х | х | х | х | х | х | х | x | х | х | х | х |
| PHU.00124 | х | х | х | х | х | х | х | х | х | x | х | х | х | х |
| PHU.00125 | х | х | х | X | х | х | х | х | х | x | х | х | х | х |
| ••• | х | х | х | X | х | х | х | х | х | x | х | х | х | х |
| Statistics | | | | | | | | | | | | | | |
| N <sup>b</sup> | х | х | х | X | х | х | х | х | х | x | х | х | х | х |
| Mean | х | х | х | X | х | х | х | х | х | x | х | х | х | х |
| SD | х | х | х | х | х | х | х | х | х | x | х | х | х | х |
| GM | х | х | х | х | х | х | х | х | х | x | х | х | х | х |
| CV % | х | х | х | х | х | х | х | х | х | X | х | х | х | Х |
| Min | х | х | х | х | х | х | х | х | х | X | х | х | х | Х |
| Max | х | х | X | х | X | х | х | X | X | X | х | х | х | х |

<sup>&</sup>lt;sup>a</sup> Times are relative to time of dosing.

Note: Samples that were collected substantially outside of the protocol-defined window are excluded from summary statistics (but not from NCA) and are indicated by an asterisks (\*).

Number of data points used to compute the summary statistics. For calculation of summary statistics, BQL values were imputed as 0 if they did not come after a PK sample concentration that is above the LLOQ and treated as missing otherwise.

Table 36: Summary Statistics for Rezafungin PK Parameters in Plasma – SAD 10 mg Dose Group

| | PK Parameters | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Statistic | C <sub>max</sub><br>(ng/mL) | T <sub>max</sub> (h) | AUC <sub>0-last</sub><br>(h*ng/mL) | AUC <sub>0-inf</sub><br>(h*ng/mL) | λz<br>(1/h) | t <sub>1/2</sub> (h) | CL/F<br>(L/h) | V <sub>z</sub> /F<br>(L) |
| N | Х | х | X | X | х | х | X | X |
| Mean | Х | х | X | X | х | х | X | X |
| SD | X | X | x | X | x | Х | X | х |
| Min | Х | х | X | X | х | Х | Х | Х |
| Median | Х | х | X | X | х | х | X | X |
| Max | Х | х | X | X | х | Х | Х | Х |
| CV % | Х | х | X | X | х | Х | Х | Х |
| GM | Х | X | x | X | x | Х | X | х |

# **APPENDIX 2. FIGURE MOCK-UPS**

# LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 66 |
|---|---|---|
| Figure 2: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group and Severity | 67 |
| Figure 3: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Any Symptoms | 68 |
| Figure 4: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Pain | 69 |
| Figure 5: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Tenderness | 69 |
| Figure 6: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Pruritus (Itching) | 69 |
| Figure 7: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Ecchymosis (Bruising), Functional Grade | 69 |
| Figure 8: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Ecchymosis (Bruising), Measurement Grade | 69 |
| Figure 9: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Induration (Hardness)/ Swelling, Functional Grade | 69 |
| Figure 10: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Induration (Hardness)/ Swelling, Measurement Grade | 69 |
| Figure 11: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Erythema (Redness), Functional Grade | 69 |
| Figure 12: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Erythema (Redness), Measurement Grade | 70 |
| Figure 13: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Nodule, Functional Grade | 70 |
| Figure 14: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Nodule, Measurement Grade | 70 |
| Figure 15: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Ulceration, Functional Grade | 70 |
| Figure 16: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Ulceration, Measurement Grade | 70 |

| Figure 17: | Proportions of Subjects with Related Adverse Events by Dose Group,<br>MedDRA SOC, and Severity | 71 |
|---|---|---|
| Figure 18: | Number of Related Adverse Events by Dose Group, MedDRA SOC, and Severity | 72 |
| Figure 19: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Parameter and Dose Group – Sodium | 73 |
| Figure 20: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Potassium | 74 |
| Figure 21: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Calcium | 74 |
| Figure 22: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Phosphorus | 74 |
| Figure 23: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Chloride | 74 |
| Figure 24: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Total Carbon Dioxide | 74 |
| Figure 25: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Glucose | 74 |
| Figure 26: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Blood Urea Nitrogen | 74 |
| Figure 27: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Creatinine | 74 |
| Figure 28: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Protein | 75 |
| Figure 29: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Albumin | 75 |
| Figure 30: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Creatine Phosphokinase | 75 |
| Figure 31: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Aspartate Aminotransferase | 75 |
| Figure 32: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Alanine Aminotransferase | 75 |
| Figure 33: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Alkaline Phosphatase | 75 |
| Figure 34: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Total Bilirubin | 75 |
| Figure 35: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Direct Bilirubin | 75 |

| Figure 36: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Hemoglobin |
|---|---|
| Figure 37: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Hematocrit |
| Figure 38: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group, – Red Blood Cell Count76 |
| Figure 39: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group –White Blood Cell Count |
| Figure 40: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Neutrophil Count |
| Figure 41: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Lymphocyte Count |
| Figure 42: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Monocyte Count |
| Figure 43: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Eosinophil Count |
| Figure 44: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Basophil Count |
| Figure 45: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Platelets |
| Figure 46: | Coagulation Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Prothrombin Time |
| Figure 47: | Coagulation Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Activated Partial Thromboplastin Time |
| Figure 48: | Coagulation Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Prothrombin International Normalized Ratio |
| Figure 49: | Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Systolic Blood Pressure |
| Figure 50: | Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Diastolic Blood Pressure |
| Figure 51: | Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Heart Rate |
| Figure 52: | Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Respiration Rate |
| Figure 53: | Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Temperature |

| Figure 54: | ECG by Scheduled Visits: Change from Baseline by Parameter – PR Interval | 81 |
|---|---|---|
| Figure 55: | ECG by Scheduled Visits: Change from Baseline by Parameter – QRS Duration | 81 |
| Figure 56: | ECG by Scheduled Visits: Change from Baseline by Parameter – QT Interval | 82 |
| Figure 57: | ECG by Scheduled Visits: Change from Baseline by Parameter – QTcF Interval | 82 |
| Figure 58: | ECG by Scheduled Visits: Change from Baseline by Parameter – RR Interval | 82 |
| Figure 59: | ECG by Scheduled Visits: Change from Baseline by Parameter –Ventricular Rate | 82 |
| Figure 60: | Individual Rezafungin Concentration within 144 h Post-Dose in Plasma Profiles – SAD 10 mg Dose Group | 83 |
| Figure 61: | Semi-Log Individual Rezafungin Concentration within 144 h Post-Dose in Plasma Profiles – SAD 10 mg Dose Group | 84 |
| Figure 62: | Individual Rezafungin Concentration for All Time Points in Plasma Profiles – SAD 10 mg Dose Group | 85 |
| Figure 63: | Semi-Log Individual Rezafungin Concentration for All Time Points in Plasma Profiles – SAD 10 mg Dose Group | 86 |
| Figure 64: | Mean Rezafungin Concentration within 144 h Post-Dose in Plasma Profiles – SAD 10 mg Dose Group | 87 |
| Figure 65: | Semi-Log Mean Rezafungin Concentration within 144 h Post-Dose in Plasma Profiles – SAD 10 mg Dose Group | 88 |
| Figure 66: | Mean Rezafungin Concentration for All Time Points in Plasma Profiles – SAD 10 mg Dose Group | 89 |
| Figure 67: | Semi-Log Mean Rezafungin Concentration for All Time Points in Plasma Profiles – SAD 10 mg Dose Group | 90 |

#### 10.1 Disposition of Subjects

### Figure 1: CONSORT Flow Diagram

[Implementation Note: CONSORT diagram will show numbers of subjects screened and enrolled, and by Dose Group will show number randomized, treated, and completed per protocol. Additionally, it will show the number of subjects excluded from analysis populations by reason for exclusion.]

This is a place holder for Figure 1. The specifications for Figure 1 are in the implementation note.
### 14.3.1.1 Solicited Reactogenicity Symptoms

# Figure 2: Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group and Severity

[Implementation Note: All local reactogenicity symptoms will be listed using consistent symptom names as the solicited reactogenicity table shells, including "Any Symptoms"]



Figure 3: Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Any Symptoms

[Implementation Note: Maximum severity on Day 1 will be calculated based on all time points collected on Day 1 (Day 1, 1 h Post-Dose and Day 1, 4 h Post-Dose). Maximum severity on Day 14 and Final Visit will be calculated based on records in memory aid and in clinic assessments. ]



| Figure 4: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Pain |
|---|---|
| | This figure will repeat Figure 3 for Pain |
| Figure 5: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Tenderness |
| | This figure will repeat Figure 3 for Tenderness |
| Figure 6: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Pruritus (Itching) |
| | This figure will repeat Figure 3 for Pruritus (Itching) |
| Figure 7: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Ecchymosis (Bruising), Functional Grade |
| | This figure will repeat Figure 3 for Ecchymosis (Bruising), Functional Grade |
| Figure 8: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Ecchymosis (Bruising), Measurement Grade |
| | This figure will repeat Figure 3 for Ecchymosis (Bruising), Measurement Grade |
| Figure 9: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Induration (Hardness)/ Swelling, Functional Grade |
| | This figure will repeat Figure 3 for Induration (Hardness)/ Swelling, Functional Grade |
| Figure 10: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Induration (Hardness)/ Swelling, Measurement Grade |
| | This figure will repeat Figure 3 for Induration (Hardness)/ Swelling, Measurement Grade |
| Figure 11: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time |

This figure will repeat Figure 3 for Erythema (Redness), Functional Grade

Point, and Severity - Erythema (Redness), Functional Grade

| Figure 12: | Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time |
|---|---|
| | Point, and Severity – Erythema (Redness), Measurement Grade |

This figure will repeat Figure 3 for Erythema (Redness), Measurement Grade

# Figure 13: Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Nodule, Functional Grade

This figure will repeat Figure 3 for Nodule, Functional Grade

# Figure 14: Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Nodule, Measurement Grade

This figure will repeat Figure 3 for Nodule, Measurement Grade

# Figure 15: Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Ulceration, Functional Grade

This figure will repeat Figure 3 for Ulceration, Functional Grade

# Figure 16: Proportions of Subjects with Solicited Reactogenicity Symptoms by Dose Group, Time Point, and Severity – Ulceration, Measurement Grade

This figure will repeat Figure 3 for Ulceration, Measurement Grade

#### 14.3.1.2 Unsolicited Adverse Events

# Figure 17: Proportions of Subjects with Related Adverse Events by Dose Group, MedDRA SOC, and Severity

[Implementation Note: This figure includes serious and non-serious unsolicited adverse events deemed related to study product. Note that this figure will present the number of subjects with types of adverse events, and a subject may not be counted more than once for the same type of adverse event but will be counted only once for the maximum severity of the respective type. Each figure panel will show counts for all SOCs observed in any Dose Group during the study (as a related AE). If the number of SOCs is too large to fit if using 2 rows of panels, then this figure will be split into multiple figures in the CSR, with 1 row of 2 panels in each figure. SOCs will be ordered alphabetically.]



### Figure 18: Number of Related Adverse Events by Dose Group, MedDRA SOC, and Severity

[Implementation Note: This figure includes serious and non-serious unsolicited adverse events deemed related to study product. Note that this figure will present total counts of adverse events, and a subject may be represented by more than one count for the same type of adverse event. Each figure panel will show counts for all SOCs observed in any Dose Group during the study (as a related AE). If the number of SOCs is too large to fit if using 2 rows of panels, then this figure will be split into multiple figures in the CSR, with 1 row of 2 panels in each figure. SOCs will be ordered alphabetically.]



## 14.3.5 Displays of Laboratory Results

## 14.3.5.1 Chemistry Results

Figure 19: Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Parameter and Dose Group – Sodium



| Figure 20: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Potassium |
|---|---|
| | This figure will repeat Figure 19 for Potassium. |
| Figure 21: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Calcium |
| | This figure will repeat Figure 19 for Calcium. |
| Figure 22: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Phosphorus |
| | This figure will repeat Figure 19 for Phosphorus. |
| Figure 23: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Chloride |
| | This figure will repeat Figure 19 for Chloride. |
| Figure 24: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Total Carbon Dioxide |
| | This figure will repeat Figure 19 for Total Carbon Dioxide. |
| Figure 25: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Glucose |
| | This figure will repeat Figure 19 for Glucose. |
| Figure 26: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Blood Urea Nitrogen |
| | This figure will repeat Figure 19 for Blood Urea Nitrogen. |
| Figure 27: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Creatinine |
| | This figure will repeat Figure 19 for Creatinine. |

| Figure 28: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Protein |
|---|---|
| | This figure will repeat Figure 19 for Protein. |
| Figure 29: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Albumin |
| | This figure will repeat Figure 19 for Albumin. |
| Figure 30: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Creatine Phosphokinase |
| | This figure will repeat Figure 19 for Creatine Phosphokinase. |
| Figure 31: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Aspartate Aminotransferase |
| | This figure will repeat Figure 19 for Aspartate Aminotransferase. |
| Figure 32: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Alanine Aminotransferase |
| | This figure will repeat Figure 19 for Alanine Aminotransferase. |
| Figure 33: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Alkaline Phosphatase |
| | This figure will repeat Figure 19 for Alkaline Phosphatase. |
| Figure 34: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Total Bilirubin |
| | This figure will repeat Figure 19 for Total Bilirubin. |
| Figure 35: | Chemistry Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Direct Bilirubin |
| | This figure will repeat Figure 19 for Direct Bilirubin. |

| | | L202 |
|---|---|---|
| 14.3.5.2 | Hematology Results | |
| Figure 36: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Hemoglobin | |
| | This figure will repeat Figure 19 for Hemoglobin. | |
| Figure 37: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Hematocrit | |
| | This figure will repeat Figure 19 for Hematocrit. | |
| Figure 38: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group, – Red Blood Cell Count | |
| | This figure will repeat Figure 19 for Red Blood Cell Count. | |
| Figure 39: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group –White Blood Cell Count | |
| | This figure will repeat Figure 19 for White Blood Cell Count. | |
| Figure 40: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Neutrophil Count | |
| Figure 40: | • | |
| | Laboratory Parameter and Dose Group – Neutrophil Count | |
| | Laboratory Parameter and Dose Group – Neutrophil Count This figure will repeat Figure 19 for Neutrophil Count. Hematology Laboratory Results by Scheduled Visits: Change from Baseline by | |
| Figure 40: Figure 41: Figure 42: | Laboratory Parameter and Dose Group – Neutrophil Count This figure will repeat Figure 19 for Neutrophil Count. Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Lymphocyte Count | |

| Figure 43: | Hematology Laboratory Results by Scheduled Visits: Change from Baseline by |
|---|---|
| | Laboratory Parameter and Dose Group – Eosinophil Count |

This figure will repeat Figure 19 for Eosinophil Count.

# Figure 44: Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Basophil Count

This figure will repeat Figure 19 for Basophil Count.

# Figure 45: Hematology Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Platelets

This figure will repeat Figure 19 for Platelets.

### 14.3.5.3 Coagulation Results

Figure 46: Coagulation Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Prothrombin Time

This figure will repeat Figure 19 for Prothrombin Time.

Figure 47: Coagulation Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Activated Partial Thromboplastin Time

This figure will repeat Figure 19 for Activated Partial Thromboplastin Time.

Figure 48: Coagulation Laboratory Results by Scheduled Visits: Change from Baseline by Laboratory Parameter and Dose Group – Prothrombin International Normalized Ratio

This figure will repeat Figure 19 for Prothrombin International Normalized Ratio.

## 14.3.6 Displays of Vital Signs

Figure 49: Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Systolic Blood Pressure



| Figure 50: | Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups | s – |
|---|---|---|
| | Diastolic Blood Pressure | |

This figure will repeat Figure 49 for Diastolic Blood Pressure.

# Figure 51: Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Heart Rate

This figure will repeat Figure 49 for Heart Rate.

# Figure 52: Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Respiration Rate

This figure will repeat Figure 49 for Respiration Rate.

# Figure 53: Vital Signs by Scheduled Visits: Change from Baseline by Parameter and Dose Groups – Temperature

This figure will repeat Figure 49 for Temperature.

## 14.3.7 Displays of ECG Measurements

Figure 54: ECG by Scheduled Visits: Change from Baseline by Parameter – PR Interval



Figure 55: ECG by Scheduled Visits: Change from Baseline by Parameter – QRS Duration

This figure will repeat Figure 54 for QRS Duration.

### Figure 56: ECG by Scheduled Visits: Change from Baseline by Parameter – QT Interval

This figure will repeat Figure 54 for QT Interval.

### Figure 57: ECG by Scheduled Visits: Change from Baseline by Parameter – QTcF Interval

This figure will repeat Figure 54 for QTcF Interval.

### Figure 58: ECG by Scheduled Visits: Change from Baseline by Parameter – RR Interval

This figure will repeat Figure 54 for RR Interval.

## Figure 59: ECG by Scheduled Visits: Change from Baseline by Parameter – Ventricular Rate

This figure will repeat Figure 54 for Ventricular Rate.

Figure 60: Individual Rezafungin Concentration within 144 h Post-Dose in Plasma Profiles – SAD 10 mg Dose Group



Figure 61: Semi-Log Individual Rezafungin Concentration within 144 h Post-Dose in Plasma Profiles – SAD 10 mg Dose Group



Figure 62: Individual Rezafungin Concentration for All Time Points in Plasma Profiles – SAD 10 mg Dose Group



Figure 63: Semi-Log Individual Rezafungin Concentration for All Time Points in Plasma Profiles – SAD 10 mg Dose Group



Figure 64: Mean Rezafungin Concentration within 144 h Post-Dose in Plasma Profiles – SAD 10 mg
Dose Group



Figure 65: Semi-Log Mean Rezafungin Concentration within 144 h Post-Dose in Plasma Profiles – SAD 10 mg Dose Group



Figure 66: Mean Rezafungin Concentration for All Time Points in Plasma Profiles – SAD 10 mg
Dose Group



Figure 67: Semi-Log Mean Rezafungin Concentration for All Time Points in Plasma Profiles – SAD 10 mg Dose Group



## APPENDIX 3. LISTINGS MOCK-UPS

# LISTINGS

| Listing 1: | 16.1.6: Listing of Subjects Receiving Investigational Product | 93 |
|---|---|---|
| Listing 2: | 16.2.1: Early Terminations or Discontinued Subjects | 94 |
| Listing 3: | 16.2.2.1: Subject-Specific Protocol Deviations | 95 |
| Listing 4: | 16.2.2.2: Non-Subject-Specific Protocol Deviations | 96 |
| Listing 5: | 16.2.3: Subjects Excluded from Analysis Populations | 97 |
| Listing 6: | 16.2.4.1: Demographic Data | 98 |
| Listing 7: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | 99 |
| Listing 8: | 16.2.5: Compliance and/or Drug Concentration Data | 100 |
| Listing 9: | 16.2.7.2: Solicited Reactogenicity Events – Local Symptoms | 101 |
| Listing 10: | 16.2.7.3: Unsolicited Adverse Events | 102 |
| Listing 11: | 16.2.8.1: Clinical Laboratory Results – Chemistry | 103 |
| Listing 12: | 16.2.8.2: Clinical Laboratory Results – Hematology | 104 |
| Listing 13: | Clinical Laboratory Results – Coagulation | 104 |
| Listing 14: | 16.2.8.3: Clinical Laboratory Results – Urinalysis | 105 |
| Listing 15: | Clinical Laboratory Results – Serology | 106 |
| Listing 16: | Screening Laboratory Results – Urine Toxicology | 107 |
| Listing 17: | Laboratory Results – Serum hCG and Pregnancy Tests | 108 |
| Listing 18: | 16.2.9.1: Vital Signs | 109 |
| Listing 19: | 16.2.9.2: Physical Exam Findings | 110 |
| Listing 20: | Listing of ECG Interval Measurements | 111 |
| Listing 21: | Listing of ECG Overall Interpretation and Comments | 112 |
| Listing 22: | Listing of ECG Findings | 113 |
| Listing 23: | Prior Medications. | 114 |
| Listing 24: | 16.2.10: Concomitant Medications | 115 |
| Listing 25: | 16.2.11.1: Pregnancy Reports – Maternal Information | 116 |
| Listing 26: | 16.2.11.2: Pregnancy Reports – Gravida and Para | 116 |
| Listing 27: | 16.2.11.3: Pregnancy Reports – Live Birth Outcomes | 117 |
| Listing 28: | 16.2.11.4: Pregnancy Reports – Still Birth Outcomes | 117 |

| _ | 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 117 |
|---|---|---|
| Listing 30: | Birth Control Listing | 118 |
| Listing 31: | Subject Level Drug Concentrations | 119 |
| Listing 32: | Subject-Specific PK Parameters | 120 |

## Listing 1: 16.1.6: Listing of Subjects Receiving Investigational Product

(This is a placeholder for the abbreviated CSR)

## 16.2 Database Listings by Subject

## **16.2.1 Discontinued Subjects**

## **Listing 2:** 16.2.1: Early Terminations or Discontinued Subjects

[Implementation Note: Category will be either "Early Termination" or "Treatment Discontinuation." In the "Reason" column, concatenate any "specify" fields, including AE number and DV number. Sort order: Dose Group, Subject ID, Category (in the case a subject both terminates early and discontinues treatment).]

| Dose Group | Subject ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Early Termination | Lost to Follow-up | 7 |

#### **16.2.2 Protocol Deviations**

## **Listing 3:** 16.2.2.1: Subject-Specific Protocol Deviations

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Subject refusal." Sort order: Dose Group, Subject ID, DV Number. If deviation resulted in AE or subject termination, or affected product stability, indicate which of those events occurred in the listing row, since columns for those 3 events were concatenated to save space.]

| Dose Group | Subject ID | DV Number | Deviation | Deviation<br>Category | Study Day | Reason for<br>Deviation | Deviation Resulted in AE or Subject<br>Termination, or Affected Product Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

## Listing 4: 16.2.2.2: Non-Subject-Specific Protocol Deviations

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Subject refusal." Sort order: Start Date, Deviation.]

| Start Date | Deviation | End Date | Reason for<br>Deviation | Deviation Resulted in Subject Termination? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|

## 16.2.3 Subjects Excluded from the Efficacy Analysis

### **Listing 5:** 16.2.3: Subjects Excluded from Analysis Populations

[Implementation Note: This data in this listing should be congruent with the "Analysis Populations by Dose Group" table. If subject not excluded from any analysis population, the subject will not appear in the listing. If the subject is excluded from multiple analysis populations, they will have one row per analysis population excluded from in the listing.

Sort order: Dose Group, Subject ID, Analysis from which Subject is Excluded (order: Safety, PK Analysis Population, PK Analysis Subset).]

| Dose Group | Subject ID | Analysis from which Subject is Excluded | Results Available? | Reason Subject Excluded | Reason Subject Excluded Specification |
|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | PK Analysis Subset | Yes | Has protocol deviations that potentially impact PK | Subject consumed food 1 hour prior to dosing |
| Note: "Ves" in the "Desults | Note: "Ves" in the "Pasults available" column indicates that available data were removed from the analysis "No" indicates that no data were available for inclusion in the analysis | | | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

## 16.2.4 Demographic Data

## Listing 6: 16.2.4.1: Demographic Data

[Implementation Note: If a subject is multi-racial, in "Race" column, note "Multiple: (list races, separated by a comma)."

Sort order: Dose Group, Subject ID.]

| Dose Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Race | Weight at Screening (kg) | Height at Screening (cm) | BMI at Screening (kg/m²) |
|---|---|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Female | 24 | Not Hispanic | Black or African American | xx | xxx | XX |

## Listing 7: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

[Implementation Note: "Condition Start Day" and "Condition End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). Rather than use exact study days, categorize as follows:

- 5 years prior to enrollment
- 1-5 years prior to enrollment
- 1-12 months prior to enrollment
- Within 1 month of enrollment
- During study
- If ongoing, display "Ongoing" in the "Condition End Day" column
- Within 1 month of enrollment
- During study
- If ongoing, display "Ongoing" in the "Condition End Day" column

It may be appropriate to add another category, based on exclusion criteria that restrict conditions within a particular time period (e.g., within 3 years prior to enrollment). In the CSR, Subject ID should be USUBJID (not PATID) for purposes of de-identification.

Sort order: Dose Group, Subject ID, MH Number.]

| Dose Group | Subject ID | <b>Medical History Number</b> | Medical History Term | MedDRA System Organ Class | MedDRA Preferred Term | <b>Condition Start Day</b> | Condition End Day |
|---|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | 1 | NUT ALLERGY | IMMUNE SYSTEM DISORDERS | FOOD ALLERGY | >5 years prior to enrollment | Ongoing |

## 16.2.5 Compliance and/or Drug Concentration Data (if available)

## Listing 8: 16.2.5: Compliance and/or Drug Concentration Data

[Implementation Note: If not dosed according to protocol, details will be given in the Comments column (manually written, not programmed). If Dose is inapplicable for subject, the date and time columns for those doses will be "N/A" and for planned doses that did not occur the date and time columns for those doses will be "not dosed."

Sort order: Dose Group, Subject ID, Dose Date, Dose Time]

| Dose Group | Subject ID | Dosed According to Protocol? | Dose Date | Dose Time | Comments |
|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Yes | ddMMMyyyy | hh:mm | |

### 16.2.7 Adverse Events

## **Listing 9:** 16.2.7.2: Solicited Reactogenicity Events – Local Symptoms

[Implementation Note: Functional grade will be displayed under "Functional Grade" column and measurement and measurement grade will be displayed together in "Measurement (Grade)" column ex: 30 (Mild)

Sort order: Dose Group, Subject ID, Time Point]

| Dose Group | Subject ID | Time Point | Assessmenta | Location | Symptom | Functional Grade | Measurement (Grade) |
|---|---|---|---|---|---|---|---|
| | | | Clinic | Upper Left | Pain | Mild | 30 (Mild) |
| | | | MA | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Reactogenicity Events eCRF. Clinic = Data collected by clinic staff during symptom assessment.

## **Listing 10:** 16.2.7.3: Unsolicited Adverse Events

[Implementation Note: If the event is ongoing (no stop date), indicate "ongoing" in the "Duration" column. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon. This listing includes all unsolicited adverse events. Sort order: Dose Group, Subject ID, AE Number.]

| Adverse<br>Event | MedDRA System<br>Organ Class | MedDRA<br>Preferred Term | Study Day | Duration of<br>AE in Days | Severity | SAE? | Relationship to Study<br>Treatment<br>(Alternate Etiology) | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose Group | Dose Group: , Subject ID: , AE Number: | | | | | | | | | |
| | | | | | | | | | | 1 |
| Comments: | | | | | | | | | | |
| Dose Group | Dose Group: , Subject ID: , AE Number: | | | | | | | | | |
| Comments: | | | | | | | | | | |
### 16.2.8 Individual Laboratory Measurements

### Listing 11: 16.2.8.1: Clinical Laboratory Results – Chemistry

[Implementation Note: These listings (for hematology, chemistry, coagulation, and urinalysis) include all laboratory results, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal results, e.g., 16.2 (Mild). Results not in the reference range, but not graded as Mild, Moderate, or Severe, should have ONR shown as the Severity Grade.

Sort order: Parameter, Dose Group, Subject ID, and Time Point. Change from Baseline column will be blank for parameters that are not numerical.]

| Dose Group | Subject ID | Time Point | Date of Assessment | Sex | Laboratory Parameter (Units) | Result (Severity Grade) | Change from Baseline | Reference Range |
|---|---|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Day 2 | ddMMMyyyy | Male | Sodium (mmol/L) | 132 (Mild) | -7 | 135 -145 |

# **Listing 12:** 16.2.8.2: Clinical Laboratory Results – Hematology

| Dose Group | Subject ID | Time Point | Date of Assessment | Sex | Laboratory Parameter (Units) | Result (Severity Grade) | Change from Baseline | Reference Range |
|---|---|---|---|---|---|---|---|---|
| | | | ddMMMyyyy | | | | | |

# **Listing 13:** Clinical Laboratory Results – Coagulation

| Dose Group | Subject ID | Time Point | Date of Assessment | Laboratory Parameter (Units) | Result (Severity Grade) | Change from Baseline | Reference Range |
|---|---|---|---|---|---|---|---|
| | | | ddMMMyyyy | | | | |

# **Listing 14:** 16.2.8.3: Clinical Laboratory Results – Urinalysis

[Implementation Notes: If parameter is determined using multiple methods, present the result from each method as a separate row, with Dipstick results preceding Complete UA results.]

| Dose Group | Subject ID | Time Point | Date of Assessment | Sex | Laboratory Parameter (Units) | Result (Severity Grade) | Reference Range |
|---|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Day 2 | ddMMMyyyy | Male | Total Protein by Dipstick | Positive (ONR) | Negative |
| SAD 1 mg | PHU.00123 | Day 2 | | Male | RBC Count by Microscopic Evaluation (/HPF) | 5 (Mild) | <5 |

## **Listing 15:** Clinical Laboratory Results – Serology

[Implementation Note: Listing will be sorted by Dose Group, Subject ID, then by Visit (order: Screening, then Unscheduled). If there are results for urine toxicology tests on an Unscheduled visit, the Study Day will be included in parentheses for the Visit.]

| Dose Group | Subject ID | Visit | HIV Antibodies | HCV Antibodies | HBsAg |
|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Screening | Negative | Negative | Negative |
| SAD 1 mg | PHU.00123 | Unscheduled (Day 4) | Negative | Negative | Negative |

### **Listing 16:** Screening Laboratory Results – Urine Toxicology

[Implementation Note: Listing will be sorted by Dose Group, Subject ID, then by Visit (order: Screening, then Unscheduled). If there are results for urine toxicology tests on an Unscheduled visit, the Study Day will be included in parentheses for the Visit.]

| Dose Group | Subject ID | Visit | Cannabinoids | Amphetamines | Barbiturates | Cocaine | Opiates | Benzodiazepines | Phencyclidine | Alcohol | Cotinine |
|---|---|---|---|---|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Screening | Negative | Negative | Negative | Negative | Negative | Negative | Negative | | |
| SAD 1 mg | PHU.00123 | Admission | Negative | Negative | Negative | Negative | Negative | Negative | Negative | | |
| SAD 1 mg | PHU.00123 | Unscheduled (Day 4) | Negative | Negative | Negative | Negative | Negative | Negative | Negative | | |

#### Listing 17: Laboratory Results - Serum hCG and Pregnancy Tests

[Implementation Note: Listing will be sorted by Dose Group, Subject ID, then by Visit (order: Screening, then Admission, then Unscheduled). If there are results for serum hCG or serum/urine pregnancy tests on an Unscheduled visit, the Study Day will be included in parentheses for the Visit. FSH testing results, if obtained, will be shown in this listing.]

| Dose Group | Subject ID | Visit | Serum HCG Result | FSH Test Result |
|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Screening | Negative | ND |
| Note: ND = Test not performed | | | | |

### 16.2.9 Vital Signs and Physical Exam Findings

### Listing 18: 16.2.9.1: Vital Signs

[Implementation Note: This listing includes all vital sign assessments, scheduled and unscheduled. All height, weight, and BMI measurements will be included in this listing as well. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal assessments, e.g., 100.7 (Mild). Sort order: Dose Group, Subject ID, Parameter, Date of Assessment, and Time of Assessment.]

| Dose Group | Subject ID | Parameter (units) | Time Point | Date of Assessment | Time of Assessment | Result (Severity Grade) | Change from Baseline | Reason for Repeat |
|---|---|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Systolic Blood Pressure (mmHg) | Day 1, 30 minutes<br>Post-Dose | ddMMMyyyy | hh:mm | 142 (Mild) | +10 | |

### Listing 19: 16.2.9.2: Physical Exam Findings

[Implementation Note: This listing includes all physical exam findings, scheduled and unscheduled. If a subject does not have any findings upon examination, they will not be included in this listing. If reported as an AE, display "Yes" with the AE Number in parentheses, e.g., "Yes (RASH, 007)". In the CSR, Subject ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Dose Group, Subject ID, Date of Assessment, Time of Assessment, Body System, and Finding.]

| Dose Group | Subject ID | Time Point | Date of Assessment | Time of Assessment | Body System | Abnormal Findings | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|---|---|---|

### 16.2.10 ECG Results and Findings

### **Listing 20:** Listing of ECG Interval Measurements

[Implementation Note: This listing includes all ECG assessments, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal assessments, e.g., 100.7 (Mild). For all change from baseline, show "+" or "-" next to the change from baseline results if an increase or decrease.

Sort order: Dose Group, Subject ID, Parameter, Date of Assessment, and Time of Assessment.]

| Dose Group | Subject ID | Sex | Parameter (units) | Time Point | Date of<br>Assessment | Time of<br>Assessment | Result (Severity<br>Grade) | Change from<br>Baseline | Replicate<br>Number | Reason for<br>Repeat |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Pre-Dose | ddMMMyyyy | | | | 1 | |
| | | | | Pre-Dose | | | | | 2 | |
| | | | | Pre-Dose | | | | | 3 | |
| SAD 1 mg | PHU.00123 | Male | QTcF (msec) | Pre-Dose<br>(Baseline) | | MEDIAN | 147 | | | |
| SAD 1 mg | PHU.00123 | Male | QTcF (msec) | Day 1, 2 h<br>Post-Dose | ddMMMyyyy | hh:mm | 450 (Mild) | +25 | | |

# **Listing 21:** Listing of ECG Overall Interpretation and Comments

[Implementation Note: This listing includes all ECG assessments, scheduled and unscheduled.

Sort order: Dose Group, Subject ID, Date of Assessment, and Time of Assessment.]

| Dose Group | Subject ID | Time Point | Date of Assessment | Time of Assessment | Interpretation | Comments |
|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Day 1, 2 h Post-Dose | ddMMMyyyy | hh:mm | Abnormal, NCS | Sinus Bradycardia |
| | | | | | Abnormal, CS | |

# **Listing 22:** Listing of ECG Findings

[Implementation Note: Sort order: Dose Group, Subject ID, Date of Assessment, Time of Assessment, Category, and Finding.]

| Dose Group | Subject ID | Time Point | Date of Assessment | Time of Assessment | Category | Finding |
|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Day 1, 2 h Post-Dose | ddMMMyyyy | hh:mm | Arrhythmia | Sinus arrhythmia |

#### **16.2.10** Concomitant Medications

### **Listing 23:** Prior Medications

[Implementation Note: Include prior medications (medications with an end date prior to dosing) only. If start date is more than 30 days before enrollment then categorize as: 1-12 months prior to enrollment, 1-5 years prior to enrollment, or 5 years prior to enrollment.

Sort order: Dose Group, Subject ID, and CM Number.]

| Dose Group | Subject ID | CM Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for a condition on Medical History?<br>(MH Description; Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | 001 | BENADRYL | 1-12 months prior<br>to enrollment | 1-12 months prior<br>to enrollment | ITCHING | No | DERMATOLOGICALS<br>(ANTIPRURITICS, INCL.<br>ANTIHISTAMINES,<br>ANESTHETICS, ETC.) |

### **Listing 24:** 16.2.10: Concomitant Medications

[Implementation Note: "Medication Start Day" and "Medication End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). For medication start dates that are > 30 days prior to enrollment, rather than use exact study days, categorize as follows:

- 5 years prior to enrollment
- 1-5 years prior to enrollment
- 1-12 months prior to enrollment

If ongoing, display "Ongoing" in the "Medication End Day" column. If taken for an AE or MH, display "Yes" with the AE or MH Number in parentheses, e.g., "Yes (RASH, 007)". In the CSR, Subject ID should be USUBJID (not PATID) for purposes of de-identification.

Sort order: Dose Group, Subject ID, and CM Number.]

| Dose<br>Group | Subject ID | CM<br>Number | Medication | Medication<br>Start Day | Medication<br>End Day | Indication | Taken for an AE? (AE Description; Number) | Taken for a condition on<br>Medical History?<br>(MH Description; Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | 001 | BENADRYL | 2 | 2 | ITCHING | Yes (MACULAR RASH; 001) | No | DERMATOLOGICALS<br>(ANTIPRURITICS, INCL.<br>ANTIHISTAMINES,<br>ANESTHETICS, ETC.) |

### 16.2.11 Pregnancy Reports

### **Listing 25:** 16.2.11.1: Pregnancy Reports – Maternal Information

| Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day Corresponding to Estimated Date of Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 26: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

a Preterm Birth

b Preterm Birth

# **Listing 27:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| egnancy Fetu<br>umber Numl | ` | Fetal Distress<br>During Labor<br>and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|

### **Listing 28:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

# Listing 29: 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|

### **Listing 30:** Birth Control Listing

[Implementation Note: If subject not of child bearing potential, indicate reason subject is not of child bearing potential in parentheses in the column Child Bearing Potential. If start date is more than 30 days before enrollment then categorize, rather than use exact study days, categorize as follows: 1-12 months prior to enrollment, 1-5 years prior to enrollment, or 5 years prior to enrollment.

Sort Order: Dose Group, Subject ID, and then by Start Day.]

| Dose Group | Subject ID | Sex | Child Bearing<br>Potential | Birth Control<br>Method | Birth Control<br>Start Day | Birth Control<br>End Day |
|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | Female | Yes | Hormonal Injections | -2 | Ongoing |

#### **Listing 31:** Subject Level Drug Concentrations

[Implementation Note: Units of nominal time and actual time vary by time point and will be provided for each time rather than in the column heading. Laboratory Reported Drug Concentration will give verbatim value reported by lab (with minimal formatting, as needed) and will use a character variable such as PC.PCORRES. Analysis Drug Concentration will report the value actually used for analysis and will use a numeric variable such as ADPC.AVAL. If one or more samples are excluded from NCA, two additional columns will be provided in the PK report listing: Excluded from NCA (Yes/No) and Reason for Exclusion from NCA.

Sort order: Dose Group, Subject ID, and Actual Time.]

| Dose Group | Subject ID | Nominal Time <sup>a</sup> | Actual Time <sup>a</sup> | Laboratory Reported<br>Drug Concentration<br>(ng/mL) | Analysis Drug<br>Concentration<br>(ng/mL) | Used in λz<br>Calculations |
|---|---|---|---|---|---|---|
| SAD 1 mg | PHU.00123 | 0 | 0 | 0 | 0 | No |

<sup>&</sup>lt;sup>a</sup>Times are relative to time of previous dose.

Note: Actual Times that were outside of protocol-defined time windows are indicated by an asterisk (\*). Samples that were collected substantially outside of the protocol-defined window are excluded from summary statistics (but not from NCA) and are indicated by two asterisks (\*\*).

# **Listing 32:** Subject-Specific PK Parameters

[Implementation Note: Sort order: Dose Group and Subject ID.]

| Dose<br>Group | Subject ID | C <sub>max</sub><br>(ng/mL) | T <sub>max</sub> (h) | AUC <sub>0-last</sub><br>(h*ng/mL) | AUC <sub>0-inf</sub><br>(h*ng/mL) | λz<br>(1/h) | t <sub>1/2</sub> (h) | CL/F<br>(L/h) | V <sub>z</sub> /F<br>(L) |
|---|---|---|---|---|---|---|---|---|---|